#### The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

Title: Reporting and Analysis Plan for a randomised, placebocontrolled, double-blind (sponsor-open), segmental LPS challenge study to investigate the pharmacodynamics of GSK2798745 in healthy participantsCompound Number: GSK2798745Effective Date: 23-JUN-2018

## **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 207464
- This RAP is intended to describe the efficacy, biomarker/pharmacodynamics, safety and pharmacokinetics analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the interim analyses and Statistical Analysis Complete (SAC) deliverable.

## **RAP Author(s):**

| Approver | Date | Approval Method |
|---|---|---|
| Statistician (Respiratory, Clinical Statistics) | Not Applicable | Not Applicable |
| Senior Director (Respiratory, Clinical Pharmacology) | 20-JUN-2018 | Pharma TMF |

Copyright 2018 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# The GlaxoSmithKline group of companies

# **RAP Team Approvals:**

| Approver | Date | Approval Method |
|---|---|---|
| Project Physician Lead (Respiratory TAU) | 20-JUN-2018 | Email |
| Clinical Investigational Lead (Respiratory TAU) | 20-JUN-2018 | Pharma TMF |
| Operations Study Lead (CPSSO) | 20-JUN-2018 | Pharma TMF |
| Data Quality Lead (CPSSO) | 21-JUN-2018 | Pharma TMF |
| Translational Scientist and Biomarker<br>Representative (Respiratory TAU) | 11-JUN-2018 | Email |
| SERM Director (GCSP) | 23-JUN-2018 | Pharma TMF |

# **Clinical Statistics and Clinical Programming Line Approvals:**

| Approver | Date | Approval Method |
|----------------------------------------------|-------------|-----------------|
| Director (Respiratory, Clinical Statistics) | 21-JUN-2018 | Pharma TMF |
| Director (Respiratory, Clinical Programming) | 20-JUN-2018 | Email |

# **TABLE OF CONTENTS**

| | | | | PAGE |
|---|---|---|---|---|
| 1. | INTRO | ODUCTIO | ON | 6 |
| _ | OL IN AN | 44 DV OF | THEY PROTOCOL INFORMATION | 0 |
| 2. | | | KEY PROTOCOL INFORMATION | |
| | 2.1. | Change | es to the Protocol Defined Statistical Analysis Plan | 6 |
| | 2.2. | | Objective(s) and Endpoint(s) | |
| | 2.3. | | Design | |
| | 2.4. | Statistic | cal Analyses | 9 |
| 3. | PLAN | NED AN | ALYSES | 10 |
| | 3.1. | | Analyses | |
| | 3.2. | Final A | nalyses | 14 |
| 4. | ANAL | YSIS PO | PULATIONS | 15 |
| | 4.1. | Protoco | ol Deviations | 15 |
| 5. | CONC | | TONG FOR DATA ANALYSES AND DATA HANDLING | |
| Э. | | | IONS FOR DATA ANALYSES AND DATA HANDLING | 16 |
| | 5.1. | | Freatment & Sub-group Display Descriptors | |
| | 5.2. | Baselin | e Definitions | 17 |
| | 5.3. | | nation of Covariates, Other Strata and Subgroups | |
| | | 5.3.1. | | |
| | | 5.3.2. | Examination of Subgroups | 17 |
| | 5.4. | Multiple | e Comparisons and Multiplicity | |
| | 5.5. | | Considerations for Data Analyses and Data Handling | |
| | | Conver | ntions | 17 |
| 6. | STUD | Y POPU | LATION ANALYSES | 19 |
| - | 6.1. | | ew of Planned Study Population Analyses | |
| | | | · | |
| 7. | | | YNAMIC AND BIOMARKER ANALYSES | |
| | 7.1. | | / Pharmacodynamic and Biomarker Analyses | |
| | | 7.1.1. | | |
| | | 7.1.2. | | |
| | | 7.1.3. | Population of Interest | 20 |
| | | 7.1.4. | Strategy for Intercurrent (Post-Randomization) Events | |
| | | 7.1.5. | Statistical Analyses / Methods | |
| | | _ | 7.1.5.1. Statistical Methodology Specification | |
| | 7.2. | | dary Pharmacodynamic Analyses | |
| | | 7.2.1. | Endpoint / Variables | |
| | | 7.2.2. | Summary Measure | |
| | | 7.2.3. | Population of Interest | |
| | | 7.2.4. | Strategy for Intercurrent (Post-Randomization) Events | |
| | | 7.2.5. | Statistical Analyses / Methods | |
| | 7.0 | <b></b> | 7.2.5.1. Statistical Methodology Specification | |
| | 7.3. | | atory Pharmacodynamic and Biomarker Analyses | |
| | | 7.3.1. | Endpoint / Variables | |
| | | 7.3.2.<br>7.3.3 | Summary Measure | 27<br>28 |
| | | 1 . 1 . 7 | COMPONENT OF THE LEST | |

| | | 7.3.4.<br>7.3.5. | Statistical | or Intercurrent (Post-Randomization) Events<br>Analyses / Methods | 28 |
|---|---|---|---|---|---|
| | | | 7.3.5.1. | Blood biomarkers | |
| | | | 7.3.5.2. | BAL exploratory biomarkers | 30 |
| | | | 7.3.5.3. | Multivariate Analysis of BAL Total Protein and Total Neutrophils | 30 |
| 8. | CVEE. | TV ANIAI ' | VSES | | 24 |
| 0. | 8.1. | | | alyses | |
| | 8.2. | | | Analyses | |
| | 8.3. | | | es | |
| 9. | PHΔR | MACOKII | NETIC ANA | LYSES | 35 |
| Ο. | 9.1. | | | inetic Analyses | |
| | 0.1. | 9.1.1. | | Variables | |
| | | <b>0</b> | 9.1.1.1. | Drug Concentration Measures | |
| | | | 9.1.1.2. | Derived Pharmacokinetic Parameters | |
| | | 9.1.2. | - | of Interest | |
| | | 9.1.3. | | Analyses / Methods | |
| | 9.2. | Seconda | | cokinetic Analyses | |
| | | 9.2.1. | | Variables | |
| | | | 9.2.1.1. | Drug Concentration Measures | |
| | | | 9.2.1.2. | Derived Pharmacokinetic Parameters | 36 |
| | | 9.2.2. | Population | of Interest | 36 |
| 10 | PHAR | MACOKII | NETIC / PH | ARMACODYNAMIC ANALYSES | 37 |
| | 10.1. | | | / Methods | |
| | | | • | | |
| 11. | REFE | RENCES | | | 38 |
| 12. | APPE | NDICES. | | | 39 |
| | 12.1. | Appendi | x 1: Protoco | ol Deviation Management and Definitions for | |
| | | | | n | 39 |
| | | 12.1.1. | Exclusions | s from Evaluable Population | 3 <mark>9</mark> |
| | 12.2. | Appendi | x 2: Schedu | lle of Activities | 40 |
| | | | | efined Schedule of Events | |
| | | 12.2.2. | | | |
| | | 12.2.3. | | period | |
| | | 12.2.4. | | Early Withdrawal | |
| | 12.3. | | | ment Windows | |
| | | 12.3.1. | | of Assessment Windows for Analyses | 45 |
| | 12.4. | | | Phases and Treatment Emergent Adverse | 16 |
| | | 12.4.1. | | Ses | |
| | | 12.4.1. | | Study Phases for Concomitant Medication | |
| | | 12.4.2. | | and LPS Emergent Flag for Adverse Events | |
| | 12.5. | | | splay Standards & Handling Conventions | |
| | 12.0. | 12.5.1. | | Process | |
| | | 12.5.1. | | Standards | |
| | | 12.5.3. | | Standards for Pharmacokinetic | |
| | 12.6. | | | I and Transformed Data | |
| | • • | | General | | |

| | 12.6.2. | Study Population | |
|---|---|---|---|
| | 12.6.3. | | |
| 12.7. | Appendix | x 7: Reporting Standards for Missing Data | 53 |
| | 12.7.1. | Premature Withdrawals | |
| | 12.7.2. | Handling of Missing Data | |
| | | 12.7.2.1. Handling of Missing and Partial Dates | <mark>5</mark> 3 |
| | | 12.7.2.2. Handling of Missing Data for Statistical | |
| | | Analysis | |
| 12.8. | Appendix | x 8: Values of Potential Clinical Importance | <mark>55</mark> |
| | 12.8.1. | Laboratory Values | 55 |
| | 12.8.2. | ECG | 56 |
| | 12.8.3. | Vital Signs | <mark>57</mark> |
| 12.9. | Appendix | x 9: Pharmacokinetic / Pharmacodynamic Analyses | <mark>5</mark> 8 |
| | 12.9.1. | Pharmacokinetic / Pharmacodynamic Dataset | |
| | | Specification | <mark>5</mark> 8 |
| 12.10. | Appendix | x 10: Abbreviations & Trade Marks | 60 |
| | 12.10.1. | Abbreviations | 60 |
| | | Trademarks | |
| 12.11. | Appendix | x 11: List of Data Displays | 62 |
| | 12.11.1. | Data Display Numbering | 62 |
| | 12.11.2. | Mock Example Shell Referencing | 62 |
| | 12.11.3. | Deliverables | 62 |
| | 12.11.4. | Study Population Tables | 63 |
| | | Pharmacodynamic and Biomarker Tables | |
| | 12.11.6. | Pharmacodynamic and Biomarker Figures | 71 |
| | | Safety Tables | |
| | 12.11.8. | Pharmacokinetic Tables | 80 |
| | 12.11.9. | Pharmacokinetic Figures | 81 |
| | 12.11.10 | Pharmacokinetic / Pharmacodynamic Figures | 82 |
| | | .ICH Listings | |
| | | Non-ICH Listings | |
| 12.12. | Appendix | x 12: Example Mock Shells for Data Displays | 89 |

# 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol:

| Revision Chronology: | | |
|---|---|---|
| Original Document<br>Number:<br>2016N304618_00 | 24-OCT-2017 | Original |
| Revised Document<br>Number:<br>2016N304618_01 | 02-FEB-2018 | The primary reason for amending the protocol is to update the number of timepoints for exploratory biomarkers. The number of blood samples for exploratory biomarkers has been reduced. |
| Revised Document<br>Number:<br>2016N304618_02 | 21-MAY-18 | The protocol was amended in response to comments from the competent authority. |

# 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

There were no changes or deviations to the originally planned statistical analysis specified in the protocol (Dated: 24/OCT/2017).

# 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To investigate the effect of<br>GSK2798745 on alveolar-septal<br>barrier permeability following LPS<br>challenge in healthy participants. | <ul> <li>Baseline adjusted total protein concentration in<br/>bronchoalveolar lavage (BAL) samples at 26 h (24 h<br/>after segmental LPS challenge).</li> </ul> |
| Secondary Objectives | Secondary Endpoints |
| <ul> <li>To investigate the effect of<br/>GSK2798745 on neutrophil levels<br/>in LPS-challenged lungs.</li> </ul> | <ul> <li>Baseline adjusted total and differential cell count of<br/>neutrophils in BAL samples at 26 h (24 h after<br/>segmental LPS challenge).</li> </ul> |
| To assess the safety and tolerability of GSK2798745 in LPS-challenged, healthy participants. | <ul> <li>Adverse events (AEs), laboratory safety<br/>assessments, 12-lead electrocardiogram (ECG),<br/>physical examination, vital signs, spirometry (forced<br/>expiratory volume in 1 second [FEV1] and forced<br/>vital capacity [FVC]), faecal occult blood test (FOBT).</li> </ul> |
| To assess the pharmacokinetics<br>(PK) of GSK2798745 in plasma in<br>LPS-challenged, healthy<br>volunteers | PK parameters of GSK2798745 in plasma (including AUC (0-26) and Cmax). |
| Exploratory Objectives | Exploratory Endpoints |
| To assess concentration of<br>GSK2798745 in BAL | <ul> <li>Levels of GSK2798745 in BAL samples at 2h and 26h<br/>after dosing</li> </ul> |

| Objectives | Endpoints |
|---|---|
| To investigate the effect of GSK2798745 on exploratory markers of endothelial barrier permeability and/or injury, and inflammation, in LPS-challenged lungs. | Baseline adjusted levels of exploratory biomarkers in blood and/or BAL. |
| To possibly assess metabolite<br>GSK3526876 (major metabolite of<br>GSK2798745) in plasma and BAL<br>samples. | Plasma and BAL concentrations of metabolite<br>GSK3526876. |
| To compare the PK of<br>GSK2798745 with the effect of<br>prophylactic dosing on alveolar-<br>septal barrier permeability<br>following LPS challenge in healthy<br>volunteers. | Comparison of PK parameters of GSK2798745 in<br>plasma and BAL with baseline corrected total protein<br>concentration in BAL. |
| To investigate the effect of<br>GSK2798745 on white blood cell<br>levels (except neutrophils) in<br>LPS-challenged lungs | Baseline adjusted total and differential cell count of<br>white blood cells (except neutrophils) in BAL<br>samples at 26 h (24 h after segmental LPS<br>challenge). |

## 2.3. Study Design



## 2.4. Statistical Analyses

The primary study objective is to investigate the effect of GSK2798745 relative to placebo on BAL total protein at 26 h post first dose (24 hours after segmental LPS challenge). In this study a Bayesian framework will be used (with non-informative priors on all model parameters) to estimate the posterior probability of any mean percentage reduction in 26 h BAL protein level (GSK2798745 relative to placebo). It is anticipated that BAL total protein will be loge transformed before model fitting. Following backtransformation treatment comparisons will be expressed as percentage changes.

### 3. PLANNED ANALYSES

## 3.1. Interim Analyses

The interim analyses will be undertaken by the study statistician and/or designates and the outputs will only be communicated to key members of the study team which may include the Project Physician Lead, Early Development Lead, Clinical Investigation Lead, Translational Biomarker Representative, Study Statistician, Project Statistician and Study Programmer(s). Following the decision made by this core group, the decision will be communicated to the wider study team. The decision will only be communicated to the site if the decision is made to stop.

The appropriate internal GSK procedures will be followed to ensure that access to unblinded participant level data is restricted to the relevant personnel performing the analysis. A secure directory will be created with restricted access for storage of data, programs, log files and outputs. Only participants contributing data towards the interim analysis will have their treatment codes unblinded as per GSK internal procedures.

Each interim analysis will be based on the predictive probability of meeting the end of study success criteria in the primary endpoint 26h BAL total protein (see Figure 2 and Table 1). An interim analysis will take place once approximately 10 participants per arm have completed the treatment period to determine whether there is sufficient rationale to continue or discontinue the study. If the decision is made to continue then a second interim analysis will occur once approximately 20 participants per arm have been recruited. Sufficient participants will be recruited to obtain up to 30 evaluable participants per arm.

Recruitment into the study will continue whilst the interim analysis is taking place unless data emerges regarding concerns about safety and tolerability. Any communication to the site regarding interim analyses will only take place if a decision to stop the study is made. Should the study be stopped, all ongoing participants will complete their treatment period whilst no further participants will be recruited into the study.

Figure 2 shows the operating characteristics that were evaluated by the study team for the chosen study design during the protocol development stage. It shows the interim analyses set-up under assumed true percentage reductions in total BAL protein for GSK2798745 relative to placebo of 0%, 15%, 30% and 50%, respectively, unconditional on variability. The schematic demonstrates all possible decision pathways the study may take. To obtain the operating characteristics of a given study design, 10,000 studies were simulated with each one taking a particular pathway and finishing in one of the pockets on the left or right of the diagram, or additional data review. The overall proportion of simulated studies reaching a particular conclusion gives the probability of a single study reaching that conclusion.

A stricter posterior probability futility threshold is implemented at the first interim to reduce the probability of incorrectly declaring futility. Furthermore, a minimum of 20 participants per arm must be recruited before declaring success. These rules are shown within the left (success) and right (futile) arrows. Under this design, assuming a true treatment effect of 30%, the overall probability of study success is approximately 83%, unconditional on variability. In addition, the probability of requiring a maximum of 20

participants per arm is approximately 61% (under the same assumption of true treatment effect of 30%). In the case of a placebo-like drug the probability of incorrectly declaring success is approximately 6% (akin to type 1 error rate). The blue boxes at the bottom of the charts show the probability that a study goes to data review, for which the results will be included as part of the headline reporting effort.

Figure 2 Interim Analysis Framework for Range of Assumed True Treatment Effects



The decision made at the interim analysis is supported by the interim predicted probability of success of the study i.e. given the treatment effect and variability observed

from the unblinded participants at the interim, the probability of the study going on to meet the predefined success criteria.

Table 1 shows the stopping criteria for interim analyses. Stopping for success is based upon the predicted probability of success (posterior probability of any percentage reduction in mean BAL total protein for GSK2798745 relative to placebo being at least 95%) whilst stopping for futility is based on the predicted probability of success or data review (posterior probability of any percentage reduction in mean BAL total protein for GSK2798745 relative to placebo being at least 75%). Note: PP = posterior probability [% reduction in mean BAL total protein for GSK2798745 relative to placebo > 0]).

| Table 1 | Success and Futility Criteria for each Interim Analysis |
|---------|---------------------------------------------------------|
|---------|---------------------------------------------------------|

| Interim<br>Analysis | Success | Futility |
|---|---|---|
| 10<br>participants<br>per arm | N/A – cannot stop for success at the first interim. | Predictive Prob ( $PP \ge 0.75$ ) $\le 0.075$ |
| 20 participants per arm | Predictive Prob (PP $\geq 0.95$ ) $\geq 0.85$ | Predictive Prob ( $PP \ge 0.75$ ) $\le 0.15$ |

## Additional analyses/outputs to support the interim analysis decision making

Because the key metric at the interim analysis is simply a probability, the key study team members will be presented with tables, summary statistics and figures for the primary analysis using the interim analysis population to help make an informed decision. Details of the planned displays provided at the interim analyses are provided in Appendix 11: List of Data Displays.

#### Technical details for calculating predictive probability of success in interim analysis

Note: The method described here is the preferred method of several ways to calculate the predictive probability of success.

The interim analyses utilise predictive inference methods to calculate the predictive probability of success. This predictive probability may be used to help determine whether there is sufficient rationale to continue/discontinue the study.

PROC MCMC in SAS (or other software offering the same methodology) will be used to sample both baseline (2 h) BAL total protein and 26 h BAL total protein (LPS lobe) from their respective interim posterior predictive distributions to generate values for predicted participants (participants yet to be recruited into the study). The number of predicted participants to be generated at the interim analysis is equal to the end of study sample size minus the interim number of participants (Equation 1). The observed and predicted participants are combined together and analysed using the primary analysis model. The end of study success criteria is then applied.

#### **Equation 1**

 $n_{predicted,j} = 30 - n_{interim,j}$ 

## where $j \in (A, P)$ indicates treatment group

There is a degree of uncertainty attached to parameters at the interim (due to the limited data) and for each iteration that fictitious participants are generated the set of predicted participants will look different, due to the random nature of simulations. Thus, to take this uncertainty into account and give an accurate representation of the predictive probability of success based on the interim data, the primary analysis is modelled 10,000 times i.e. the observed data is combined with a different simulated set of future participants 10,000 times. The proportion of primary analyses that trigger the end of study success criteria gives the predictive probability of success if the study was to continue from the interim.

Data is anticipated to require (log<sub>e</sub>) transformation before modelling. Baseline will be centred after transformation to improve mixing. General steps to calculating the predictive probability of success at the interim are given here. Consult the GSK statistician for more detailed steps (including the corresponding SAS program).

1. The linear predictor will be the same as the primary analysis model (assuming no further covariates are included) and will include the parameters:

| Туре | Name (#Levels) | Parameters | Priors |
|---|---|---|---|
| Fixed Categorical | Intercept (1) | #1 Intercept | N(Mean=0, |
| | T | #4 Dia I | Var=1E6) |
| | Treatment (2) | #1 Placebo | N(Mean=0, |
| | | W2 2 2 1 1 2 2 2 2 2 2 2 2 2 2 2 2 2 2 2 | Var=1E6) |
| | | #2 GSK2798745 | N/a |
| Fixed Continuous | Baseline BAL total | Linear relationship | N(Mean=0, |
| | protein | between baseline | Var=1E6) |
| | | and LPS lobe 26h | |
| | | BAL total protein | |
| | | (baseline slope). | |

- 2. The standard deviation parameters will be fitted with non-informative gamma priors with shape=0.001 and scale=0.001.
- 3. Participant id numbers for future participants will be created to achieve the maximum sample size of 60 (30 per treatment group) as described by Equation 1. Predicted participants will be allocated treatment codes using study-specific treatment block size.
- 4. The data set to be passed through PROC MCMC will contain complete data for observed interim participants plus treatment and id codes for future participants (baseline (2h) and 26h total protein will be missing).
- 5. A model statement for baseline BAL total protein will be set up within PROC MCMC with a non-informative prior N(Mean=0, Var=1E6) for mean and non-informative

- prior gamma(shape=0.001, scale=0.001) for standard deviation. This allows baseline values to be sampled for future participants from the interim posterior predictive distribution that includes data for current participants.
- 6. The outpost statement will be used to create an output dataset for posterior predictive samples from each MCMC iteration.
- 7. A series of diagnostic checks will be undertaken (see Section 7.1.5.1 (model checking & diagnostics) for further details).
- 8. A series of data manipulation steps are required to merge the observed data with each of the predicted future data sets. The number of data sets is equal to the number of MCMC iterations but all should be contained within one overall data set and labelled according to which MCMC iteration the "study" belongs to.
- 9. This overall dataset will be passed into PROC MCMC fitting the same primary analysis model but without the predictions. A BY statement will fit the model separately to each dataset (made up of observed and predicted participants). A POSTSUMMARIES option will report summaries of the parameters of interest including the primary endpoint success criteria as a flag variable ( *Posterior probability* [% reduction in mean BAL total protein for GSK2798745 relative to placebo > 0 ]  $\geq$  0.95 ) as well as the probability of being within the data review region ( *Posterior probability* [% reduction in mean BAL total protein for GSK2798745 relative to placebo > 0 ]  $\geq$  0.75 ).
- 10. The proportion of complete studies (observed + predicted participants) meeting the success criteria will be computed. The proportion meeting the success criteria gives the predictive probability of success at the interim.
- 11. The predictive probability of success is compared with the criteria described in Table 1 to support the decision at the interim analysis.

# 3.2. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All participants have completed the study as defined in the protocol.
- 2. All required database cleaning activities have been completed and final database release (DBR) and database freeze (DBF) has been declared by Data Management.
- 3. All criteria for unblinding the randomization codes have been met.
- 4. Randomization codes have been distributed according to RandAll NG procedures.

### 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Screened | All participants that signed the ICF and were screened for eligibility | Study Population |
| All Subjects | <ul> <li>All randomized participants who received at least one dose of study treatment.</li> <li>This population will be based on the treatment the participant actually received.</li> </ul> | <ul><li>Study Population</li><li>Safety/tolerability</li></ul> |
| Evaluable | <ul> <li>All participants for whom results of the primary analysis can be determined i.e. all randomised participants who received two correct doses of study treatment, received LPS and saline segmental challenge (in contralateral lobes) and for which results of both baseline (2h) and LPS lobe (26h) BAL samples are evaluable.</li> <li>This population will be based on the treatment the participant actually received.</li> </ul> | <ul> <li>BAL Pharmacodynamic</li> <li>BAL Biomarker</li> <li>Blood Biomarker</li> </ul> |
| Pharmacokinetic (PK) | All participants in the All Subjects population who had at least 1 non-missing PK assessment (Non-quantifiable [NQ] values will be considered as non-missing values). | Pharmacokinetic |

Refer to Appendix 11: List of Data Displays which details the population used for each display.

#### 4.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.

Important deviations which result in exclusion from the analysis population will also be summarised and listed. (Please refer to Appendix 1: Protocol Deviation Management and Definitions for Evaluable Population).

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan Version 1.0 (Dated: 18/JUN/2018).

- Data will be reviewed prior to unblinding and freezing the database to ensure all important deviations and deviations which may lead to exclusion from the analysis are captured and categorised on the protocol deviations dataset.
- This dataset will be the basis for the summaries and listings of protocol deviations.

A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

# 5.1. Study Treatment & Sub-group Display Descriptors

| Treatment Group Descriptions | | | |
|----------------------------------------|------------|--------------|---|
| RandAll NG Data Displays for Reporting | | | |
| Code Description Description Order in | | Order in TLF | |
| Α | Placebo | Placebo | 1 |
| В | GSK2798745 | GSK2798745 | 2 |

Treatment comparisons will be displayed as follows using the descriptors as specified:

# 1. GSK2798745 vs. Placebo

| Parameter | Study Assessments Considered as Baseline | | | | Baseline | |
|---|---|---|---|---|---|---|
| | Screening<br>(Days -28 to -<br>2) | Day -1 | Day 1 Pre-<br>dose | Day 1 1h | Day 1 2h <sup>1</sup> | Used in<br>Data<br>Display |
| Pharmacodyna | mic | | | | | |
| BAL Total<br>Protein | | | | | X | Day 1 2h |
| BAL Neutrophil Count (Total and Differential) | | | | | X | Day 1 2h |
| Safety | | | | | | |
| 12-lead ECG <sup>2</sup> | Х | Χ | X | | | Day 1<br>Pre-dose |
| Vital signs<br>(blood<br>pressure,<br>heart rate) <sup>3</sup> | Х | Х | Х | Х | | Day 1<br>Pre-dose |
| Temperature | Х | Х | Х | Х | Х | Day 1<br>Pre-dose |
| Spirometry<br>(FEV1, FVC) <sup>4</sup> | | Х | Х | | | Day 1<br>Pre-dose |
| Laboratory assessments <sup>5</sup> | | Х | | | | Day -1 |
| Exploratory Bio | omarkers | | | | • | |
| BAL<br>Biomarkers | | | | | Х | Day 1 2h |

#### NOTES:

- 1. Immediately before BAL sampling/LPS challenge
- 2. Triplicate at Screening, day-1 and day 1 pre-dose. Single measurements at time points after dosing.
- 3. Blood pressure and heart rate in triplicate.
- 4. Forced expiratory volume in 1 second (FEV1) and forced vital capacity (FVC). Triplicate measurements at each time point, the highest of which should be recorded in the case report form.
- 5. Haematology, clinical chemistry (including liver chemistry), cardiac troponins, urianalysis and coagulation profile.

#### 5.2. Baseline Definitions

If the "baseline used in data display" is missing for a parameter, then the study assessment considered as a baseline closest in time to this will replace this as the baseline used in displays. If all study assessments considered as baseline are missing then no derivation will be performed and baseline will be set to missing.

## 5.3. Examination of Covariates, Other Strata and Subgroups

#### 5.3.1. Covariates and Other Strata

The list of covariates and other strata may be used in descriptive summaries and statistical analyses, some of which may also be used for subgroup analyses. Additional covariates and other strata of clinical interest may also be considered.

| Category | Details |
|------------|--------------------------------------------------------------|
| Covariates | Baseline (2h) total protein, 26h total protein (saline lobe) |

#### NOTES:

The covariates listed are those that may be used in analyses.

The default statistical model for BAL markers is to fit an analysis of covariance (ANCOVA) model with baseline (2h BAL) response and treatment group as covariates and 26h BAL response as the response variable. Additional covariates with the use of clinical expertise and statistical tools (raw plots and model selection criteria) may be considered such as age and gender.

#### 5.3.2. Examination of Subgroups

There are no planned subgroup analyses.

# 5.4. Multiple Comparisons and Multiplicity

Due to the extensive use of a Bayesian framework and the early phase/exploratory nature of this study there will be no explicit multiplicity adjustments. Moreover, the decision framework for study success/fail is predetermined.

# 5.5. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---------|----------------------------------------------------------------|
| 12.3 | Appendix 3: Assessment Windows |
| 12.4 | Appendix 4: Study Phases and Treatment Emergent Adverse Events |
| 12.5 | Appendix 5: Data Display Standards & Handling Conventions |
| 12.6 | Appendix 6: Derived and Transformed Data |
| 12.7 | Appendix 7: Reporting Standards for Missing Data |
| 12.8 | Appendix 8: Values of Potential Clinical Importance |

# 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the All Subjects population, unless otherwise specified.

Study population analyses including analyses of participants' disposition, protocol deviations, demographic and baseline characteristics, prior and concomitant medications, and exposure and treatment compliance will be based on GSK Core Data Standards. Details of the planned displays are presented in Appendix 11: List of Data Displays.

## 7. PHARMACODYNAMIC AND BIOMARKER ANALYSES

## 7.1. Primary Pharmacodynamic and Biomarker Analyses

#### 7.1.1. Endpoint / Variables

The primary endpoint is defined as BAL total protein (in the lobe in which LPS was administered) at 26h post first dose (24 hours after segmental LPS challenge). A Bayesian framework will be used (with non-informative priors on all model parameters) to estimate the posterior probability of any percentage reduction in mean 26 h BAL protein level (GSK2798745 relative to placebo). It is anticipated that BAL total protein will be loge transformed to improve normality before model fitting. Following back-transformation treatment comparisons will be expressed as percentage changes. Details of data transformations are described in Appendix 6: Derived and Transformed Data.

## 7.1.2. Summary Measure

Following back-transformation, treatment comparison will be expressed as an adjusted median posterior percentage reduction in 26h total protein level for GSK2798745 compared to placebo, along with corresponding 95% credible interval.

## 7.1.3. Population of Interest

The primary analyses will be based on the Evaluable population.

## 7.1.4. Strategy for Intercurrent (Post-Randomization) Events

Since this is a proof of mechanism study, the estimand of interest in the primary analysis is the treatment effect (GSK2798745 c.f. placebo) for participants in the Evaluable population i.e. all randomised participants who received the two correct doses of study treatment, received LPS and saline segmental challenge (in contralateral lobes) and for which results for both baseline (2h) and 26h (LPS lobe) BAL samples are evaluable and did not have any major deviations affecting the primary endpoint. Given that the primary analyses are based on the Evaluable population in healthy participants, any intercurrent events such as treatment discontinuation will result in exclusion of the data from the analysis and no missing data imputation will occur.

## 7.1.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 11: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 7.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

## 7.1.5.1. Statistical Methodology Specification

#### **Endpoint / Variables**

- BAL total protein at 26h (LPS lobe).
- It is anticipated that pharmacodynamic and biomarker endpoints will require logetransformation in all analyses to improve the assumption of normality and hence improve model fitting. Following model fitting, back-transformation will occur and treatment effects (GSK2798745 relative to placebo) will be expressed as a percentage change.

## **Model Specification**

- The model described below is the default statistical model for BAL biomarkers with BAL samples taken at 2 h and 26 h. \*\*analyte\*\* in the text below should be replaced by the specific BAL endpoint in the analysis.
- The endpoint will be analysed using an analysis of covariance (ANCOVA) model fitted in a Bayesian framework with covariates having non-informative priors using PROC MCMC in SAS.
- The terms to be fitted in the model:

| Туре | Name |
|---|---|
| Dependent variable | BAL **analyte** at 26 h (LPS lobe) |
| Fixed continuous independent variables | Baseline (2 h) BAL **analyte** |
| Fixed categorical independent variables | Treatment (GSK2798745, Placebo) |

Information on the effects and prior distributions for parameters:

| Туре | Name (#Levels) | Parameters | Priors |
|---|---|---|---|
| Fixed Categorical | Intercept (1) | #1 Intercept | N(Mean= 0,<br>Var=1E6) |
| | Treatment (2) | #1 Placebo | N/a (constraint = 0) |
| | | #2 GSK2798745 | N(Mean=0,<br>Var=1E6) |
| Fixed Continuous | Baseline (2h) BAL **analyte** | Linear relationship<br>between baseline<br>(2 h) and 26 h LPS<br>lobe BAL<br>**analyte**<br>(baseline slope). | N(Mean=0,<br>Var=1E6) |

- The residual variance will be fitted with an non-informative inverse-gamma prior, igamma(shape=0.0001, scale=0.0001).
- Any centering of variables is to occur after any transformation. Baseline (2h) BAL \*\*analyte\*\* is to be centered to improve mixing in PROC MCMC.
- An optional exploration/model building step may take place by adding other covariates to the model that may explain a significant proportion of variance in the response and/or imbalance between treatment groups at baseline and/or be justified by biological rationale/expert

- judgment or statistical tools (raw plots and model selection criteria). Only the results of the final model would be reported in the Clinical Study Report (CSR).
- For the final model, appropriate combinations of model parameters should be combined to
  obtain treatment effects of interest, including performing any back-transformations that are
  required. For example, assuming loge transformation is required, the percentage change in 26h
  BAL \*\*analyte\*\* will be obtained by computing exp(β<sub>GSK2798745</sub>) for each MCMC iteration, which
  should be programmed between the BEGINNODATA and ENDNODATA statements (within
  PROC MCMC procedure).
- To obtain probability statements for parameters/effects of interest use binary flag variables. For
  each MCMC iteration if the condition is satisfied the iteration is flagged as a 1, if not it is
  flagged as 0. The proportion of iterations flagged as 1 gives the posterior probability of the
  statement of interest i.e. the proportion of MCMC iterations for which the percentage reduction
  in BAL \*\*analyte\*\* for GSK2798745 c.f. placebo is greater than zero.
  - $\circ$  For example, the SAS syntax for computing the flag for any percentage reduction in BAL \*\*analyte\*\* would be: flagsuccess = (ratio < 1); . Where ratio is the parameter used to store the ratio for adjusted posterior medians, GSK2798745 relative to placebo, calculated as  $exp(β_{GSK2798745})$ , and flagsuccess being the binary success/fail flag.

# **Model Checking & Diagnostics**

Ways to assess model appropriateness and fit can be assessed using a variety of tools. Some examples of methods are listed here:

- Use the DIC alongside expert judgment/biological rationale to select the most appropriate model. A difference in DIC between two models is >10 is generally considered substantial evidence of an important difference in model fit. Difference in DIC of <5 may be considered negligible.
- Examine trace plots for fixed parameters to evaluate whether there is constant mean and variance, that the chain is moving around the parameter space freely and moving rapidly between the extremes to show that the chain is stationary and mixing.
- Run at least 2 chains starting at different initial values. If all chains converge to the same point, then this is evidence of consistent convergence. Overlapping trace plots give visual reference for this. Running multiple chains is achieved by either by specifying initial values using begincnst/endcnst and using a by statement to run for each chain, or by using a macro to run PROC MCMC multiple times with initial values specified on the parms statement and different seeds specified for each run. Please consult GSK statistician for more details, including SAS syntax.
- The MCSE should be compared with the standard deviation of the posterior distribution (SD) to
  ensure that only a fraction of the posterior variability is due to simulation error. The ratio
  MCSE/SD should typically be ≤ 0.01.
- Autocorrelation plots should be used to assess the correlation between each draw and its kth lag. The further the lag from the original measure the smaller you expect the correlation to be.
- Rather than using the prior distribution to generate starting values for parameters in the model, use raw plots or PROC MIXED (frequentist equivalent to Bayesian) parameter estimates to help determine starting values. This should help the model converge quicker and reduces the number of burn-in iterations required.
- Tailor the number of burn-in iterations, thinning, starting values, number of posterior samples

(10,000 minimum) to ensure satisfactory model fitting and diagnostic plots.

 As an optional check, use residual plots from the PROC MIXED (frequentist equivalent to Bayesian) model to examine model fit (relevant because non-informative priors are used in the analysis). Residuals should be normally distributed (assessed with a histogram or normal probability plot). Residuals and fitted values should be uncorrelated (assessed by plotting against each other and should appear random with no structure). Any pattern suggests that the model is not appropriate. The same plot can be used to examine if there is constant variance.

#### **Model Results Presentation**

Point estimates (median values of posterior distributions), the standard deviation of the
posterior distribution (SDs) and 95% credible intervals (CrI) intervals will be presented for each
treatment group and treatment comparison (absolute and percentage change). A number of
posterior probability statements will also be expressed, as described in Table 2.

 Table 2
 Posterior Probability Statements of Interest

| Posterior Probability Statement (where X = treatment ratio of GSK2798745 / Pbo) | Interpretation |
|---|---|
| PP ( $X \le 0.25$ ) | Posterior probability of at least a 75% reduction in mean BAL **analyte** |
| PP ( X ≤ 0.5 ) | GSK2798745 relative to placebo Posterior probability of at least a 50% reduction in mean BAL **analyte** GSK2798745 relative to placebo |
| PP ( X ≤ 0.75 ) | Posterior probability of at least a 25% reduction in mean BAL **analyte** GSK2798745 relative to placebo |
| PP ( X ≤ 0.9 ) | Posterior probability of at least a 10% reduction in mean BAL **analyte** GSK2798745 relative to placebo |
| PP ( X ≤ 1 ) | Posterior probability of any reduction in mean BAL **analyte** GSK2798745 relative to placebo |
| PP ( X > 1) | Posterior probability of any increase in mean BAL **analyte** GSK2798745 relative to placebo |
| PP (X > 1.1) | Posterior probability of at least a 10% increase in mean BAL **analyte** GSK2798745 relative to placebo |
| PP (X > 1.25) | Posterior probability of at least a 25% increase in mean BAL **analyte** GSK2798745 relative to placebo |
| PP (X > 1.5) | Posterior probability of at least a 50% increase in mean BAL **analyte** GSK2798745 relative to placebo |
| PP (X > 1.75) | Posterior probability of at least a 75% increase in mean BAL **analyte** GSK2798745 relative to placebo |

- Point estimates for each treatment group and treatment comparison (absolute and percentage change) will be expressed graphically. See Appendix 11: List of Data Displays for example displays.
- Plots of the posterior distributions for 26 h BAL \*\*analyte\*\* (back-transformed) will be
  presented for each treatment arm. In addition, the posterior distributions for the absolute
  difference and percentage change in 26 h BAL \*\*analyte\*\* for GSK2798745 relative to placebo
  will be presented.

## Sensitivity and Supportive Analyses

- Sensitivity analysis 1: Assess whether there is a difference in baseline (2h) concentrations between treatment groups. The design of the study is such that baseline is observed 2 hours after the first dose of study treatment (see Figure 1). Thus, there is opportunity for inhibition of the TRPV4 channel and regulation of endothelial permeability before the baseline (2h) BAL is performed and instillation of LPS and saline challenges. Should there be a significant difference in baseline (2h) \*\*analyte\*\* between treatment arms this may be interpreted as initial concentrations (normal conditions) of \*\*analyte\*\* are being reduced. For example, '745 may reduce baseline BAL \*\*analyte\*\* for GSK2798745 c.f. placebo. This will be investigated through the use of a Bayesian ANOVA model with 2h \*\*analyte\*\* as the dependent variable and treatment group as the independent variable. See Appendix 11: List of Data Displays for further details.
- Sensitivity analysis 2: The primary analysis model may be fitted to include 26 h \*\*analyte\*\* (saline lobe) as a covariate. In a supportive analysis, the model will assess whether administration of saline in the contralateral lobe is associated with 26 h \*\*analyte\*\* in the lobe in which LPS and treatment are administered. If this is the case, then one explanation could be that the segmental LPS may have "spilled over" into other areas of the lungs including the saline lobe. This could also lead to a lower than anticipated LPS dose in the LPS lobe. The analysis would be supported by graphical displays of individual participants and their three lobe measurements (see Appendix 11: List of Data Displays for example displays). Secondly, a positive relationship between contralateral lobes could be interpreted as the BAL procedure resulting in some impact on the endothelial/epithelial lining i.e. the BAL procedure itself results in more irritation of the tissue and stimulates a biological response to a greater extent than anticipated and this results in increased permeability. Thus, by adjusting for 26 h BAL \*\*analyte\*\* (saline lobe) the model is partitioning any effect on BAL total protein due to the procedure and due to the LPS/study treatment. Another reason could be that saline impacts upon permeability. This list is not exhaustive and only speculates on the reasoning behind a significant impact in pulmonary edema in the saline lobe. Further clinical and biological expertise is required to draw any conclusions.
- Sensitivity analysis 3: A sensitivity analysis may be conducted to exclude participants for which their 26 h BAL \*\*analyte\*\* in the saline lobe increases by at least 40% relative to baseline. This is the 95th percentile of the credible interval for 11 participants that underwent segmental LPS challenge over 2 periods (measured at baseline and 26 h) at the Fraunhofer Institute, Germany [Holz, 2015]. The median for 26 h BAL total protein in the saline lobe was 13.7% (95% Crl 8.8%, 40.4%). This sensitivity analysis is being conducted because some participants may have received a greater dose of LPS than anticipated, be more sensitive to the LPS dose, the BAL procedure may have been more invasive than anticipated, etc. This may confound any observed treatment effect.

## 7.2. Secondary Pharmacodynamic Analyses

#### 7.2.1. Endpoint / Variables

BAL total and differential neutrophil count (in the lobe in which LPS was administered) at 26 hours. A Bayesian framework will be used (with non-informative priors) to estimate the posterior probability of any percentage reduction in median 26 h (24 h post-LPS) BAL response (GSK2798745 relative to placebo). It is anticipated that BAL analytes will be loge transformed to improve normality before model fitting. Following back-transformation treatment comparisons will be expressed as percentage changes. Details of data transformations are described in Appendix 6: Derived and Transformed Data.

## 7.2.2. Summary Measure

Following back-transformation, treatment comparison will be expressed as an adjusted median posterior percentage reduction in 26 h BAL analyte level for GSK2798745 compared to placebo, along with corresponding 95% highest posterior density interval.

## 7.2.3. Population of Interest

The secondary pharmacodynamic analyses will be based on the Evaluable population, unless otherwise specified.

#### 7.2.4. Strategy for Intercurrent (Post-Randomization) Events

See Section 7.1.4.

## 7.2.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 11: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 7.2.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

### 7.2.5.1. Statistical Methodology Specification

# **Endpoint / Variables**

- BAL total and differential neutrophil count at 26 h (LPS lobe).
- It is anticipated that pharmacodynamic and biomarker endpoints will require log-transformation in all analyses to improve the assumption of normality and hence improve model fitting.
   Following model fitting, back-transformation will occur and treatment effects (GSK2798745 relative to placebo) will be expressed as a percentage change.
- The derivation of differential cell count is given in Section 12.6.3.

# **Model Specification**

• See Section 7.1.5.1.

#### **Model Checking & Diagnostics**

• See Section 7.1.5.1.

#### **Model Results Presentation**

• See Section 7.1.5.1.

# 7.3. Exploratory Pharmacodynamic and Biomarker Analyses

### 7.3.1. Endpoint / Variables

Table 3 gives the matrices and sampling schemes for each of the exploratory biomarker endpoints.

Table 3 Exploratory Biomarkers and Corresponding Sampling Schemes

| Matrix | Endpoint / Analyte | Sampling<br>Scheme |
|---|---|---|
| BAL | Albumin | 2h, |
| DAL | | |
| | SP-D | 26h |
| | vWF | |
| | IL-6 | |
| | IL-8 | |
| | TNF-alpha | |
| | MPO | |
| | Urea | |
| | White blood cell counts and differentials (except | |
| | neutrophils) | |
| Blood | Total protein (plasma) | 2h, |
| | Albumin (plasma) | 3h, |
| | SP-D (serum) | 8h, |
| | vWF (serum) | 26h |
| | IL-6 (serum) | |
| | IL-8 (serum) | |
| | TNF-alpha (serum) | |
| | Immature SP-B (serum) | |
| | urea (plasma) | |
| | CRP (serum) | |

## 7.3.2. Summary Measure

#### **BAL Biomarkers**

Exploratory BAL biomarkers will be analysed and reported in the same manner as the primary pharmacodynamic data (without the sensitivity analyses) (refer to Section 7.1 for further details). Treatment comparison will be expressed (following back-transformation) as an adjusted median posterior percentage change for GSK2798745 compared to placebo, along with corresponding 95% credible interval.

## **Blood Biomarkers**

Treatment comparisons will be expressed (following back-transformation) as an adjusted median posterior percentage change for GSK2798745 compared to placebo at each of the sampling timepoints (2h, 3h, 8h and 26h).

## 7.3.3. Population of Interest

Analyses will be based on the Evaluable population for both the BAL biomarker and blood biomarker analyses.

#### 7.3.4. Strategy for Intercurrent (Post-Randomization) Events

See Section 7.1.4.

## 7.3.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 11: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 7.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

#### 7.3.5.1. Blood biomarkers

The following text is the general method for analysing and reporting blood biomarkers that follow the sampling scheme in Table 3.

#### **Endpoint / Variables**

- Each blood biomarker and the sampling timepoints are listed in Table 3.
- It is anticipated that biomarkers will require log-transformation in all analyses to improve model fitting. Following model fitting, back-transformation will occur and treatment comparisons at each of the sampling timepoints will be expressed as a percentage change for GSK2798745 relative to placebo.

#### **Model Specification**

- Each blood biomarker will be analysed using a repeated measures mixed model (MMRM) fitted in a Bayesian framework with all covariates having non-informative priors using PROC MCMC in SAS or other software.
- \*\*analyte\*\* in the text below should be replaced by the specific blood biomarker in the analysis.
- The terms to be fitted in the model:

| Туре | Name |
|---|---|
| Dependent variable | **analyte** response |
| Fixed categorical independent variables | <ul> <li>Treatment</li> <li>Sampling timepoint</li> <li>Sampling timepoint interacted with treatment</li> </ul> |

Information on the effects and prior distributions for parameters:

| Туре | Name (#Levels) | Parameters | Priors |
|-------------|--------------------|-------------------|---------------------|
| Fixed | Intercept (1) | #1 Intercept | N(Mean= 0, Var=1E6) |
| Categorical | Treatment (2) | #1 Placebo | N/a (constraint=0) |
| | | #2 GSK2798745 | N(Mean=0, Var=1E6) |
| | Sampling Timepoint | #1 2h | N/a (constraint=0) |
| | (4) | #2 3h | N(Mean=0, Var=1E6) |
| | | #3 8h | N(Mean=0, Var=1E6) |
| | | #4 26h | N(Mean=0, Var=1E6) |
| | Treatment*Sampling | #1 Placebo*2h | N/a (constraint=0) |
| | Timepoint (8) | #2 Placebo*3h | N/a (constraint=0) |
| | | #3 Placebo*8h | N/a (constraint=0) |
| | | #4 Placebo*26h | N/a (constraint=0) |
| | | #5 GSK2798745*2h | N/a (constraint=0) |
| | | #6 GSK2798745*3h | N(Mean=0, Var=1E6) |
| | | #7 GSK2798745*8h | N(Mean=0, Var=1E6) |
| | | #8 GSK2798745*26h | N(Mean=0, Var=1E6) |

- The default prior for the VCV matrix would be an Inverse-Wishart with parameters k and S (where S = (k p 1) \* R and p = dimension of the VCV matrix). Under this framework, R can be thought of as a best guess for the VCV of the endpoints/timepoints being modelled. Care should be taken in the choice of k and R for each endpoint to ensure it is uninformative.
- Separate variance-covariance matrices will be used for treatment groups if there is sufficient
  information/data to allow for this, i.e. convergence occurs for all parameters and values do not
  get "stuck" at zero. If there is not sufficient information then the default position is for treatment
  groups to share a common variance-covariance matrix.
- An optional exploration/model building step may take place by adding other covariates to the
  model that may explain a significant proportion of variance in the response and/or imbalance
  between treatment groups at baseline and/or be justified by biological rationale/expert
  judgment or statistical tools (raw plots and model selection criteria). Only the results of the final
  model would be reported in the Clinical Study Report (CSR).
- For the final model, appropriate combinations of model parameters should be combined to obtain treatment effects of interest, including performing any back-transformations that are required. For example, assuming loge transformation is required, the percentage change at 8h for GSK2798745 relative to placebo will be obtained by computing exp(β<sub>GSK2798745</sub> + β<sub>GSK2798745\*8h</sub> β<sub>8h</sub>) for each MCMC iteration, which should be programmed between the BEGINNODATA and ENDNODATA statements (within PROC MCMC procedure).
- To obtain probability statements for parameters/effects of interest use binary flag variables. For each MCMC iteration if the condition is satisfied the iteration is flagged as a 1, if not it is flagged as 0. The proportion of iterations flagged as 1 gives the posterior probability of the

- statement of interest i.e. the proportion of MCMC iterations for which the percentage reduction in the BAL biomarker for GSK2798745 c.f. placebo for the specified sampling timepoint is greater than zero.
- For example, the SAS syntax for computing the flag for any percentage reduction in BAL \*\*analyte\*\* would be:  $flagsuccess\_8h = (ratio\_8h < 1)$ ; . Where  $ratio\_8h$  is the parameter used to store the ratio of adjusted posterior medians for GSK2798745 relative to placebo at the 8h sampling timepoint, calculated as  $exp(\beta_{GSK2798745} + \beta_{GSK2798745*8h} \beta_{8h})$ , and  $flagsuccess\_8h$  being the binary success/fail flag.

## **Model Checking & Diagnostics**

See Section 7.1.5.1 (Model Checking and Diagnostics)

#### **Model Results Presentation**

- Point estimates (median values of posterior distributions), the standard deviation of the
  posterior distribution (SDs) and 95% credible intervals (CrI) intervals will be presented for each
  treatment group and treatment comparison (absolute and percentage change) at each
  sampling time point. A number of posterior probability statements will also be expressed, as
  described in Table 2 of Section 7.2.5.1 (Model Results Presentation) for each timepoint.
- Point estimates for each treatment group and treatment comparison (absolute and percentage change) at each timepoint will be expressed graphically. See Appendix 11: List of Data Displays for example displays.
- Plots of the posterior distributions for each timepoint (back-transformed) will be presented for each treatment arm. In addition, the posterior distributions for the absolute difference and percentage change at each timepoint for GSK2798745 relative to placebo will be presented.
- Where appropriate, LLQs and ULQs should be displayed in figures through the use of dashed horizontal lines.
- PD\_T2: The adjusted percentage change in analyte should be expressed as a reduction or increase (GSK2798745 c.f. placebo) depending on the analyte and the desired direction of treatment effect e.g. % reduction/increase GSK2798745 relative to placebo.
- PD\_F5: The adjusted percentage change in analyte should be expressed as a reduction or increase (GSK2798745 c.f. placebo) depending on the specific analyte and the desired direction of treatment effect e.g. % reduction/increase GSK2798745 relative to placebo.

#### 7.3.5.2. BAL exploratory biomarkers

The strategy for analysing and reporting BAL exploratory biomarkers will follow the same structure as the primary analysis (see Section 7.1). Details of outputs can be found in Appendix 11: List of Data Displays.

#### 7.3.5.3. Multivariate Analysis of BAL Total Protein and Total Neutrophils

This analysis may be conducted to better understand the correlation between the endpoints and will be supported by tables and figures.

### **Endpoint / Variables**

- Absolute BAL total protein and total neutrophil counts
- It is anticipated that biomarkers will require log-transformation in all analyses to improve model fitting. Following model fitting, back-transformation will occur and treatment comparisons at each of the sampling timepoints will be expressed as a percentage change for GSK2798745 relative to placebo.

#### **Model Specification**

- Each blood biomarker will be analysed using a repeated measures mixed model (MMRM) fitted in a Bayesian framework with all covariates having non-informative priors using PROC MCMC in SAS.
- \*\*analyte\*\* in the text below should be replaced by the specific blood biomarker in the analysis.
- The terms to be fitted in the model:

| Туре | Name |
|-----------------------------------------|---------------------|
| Dependent variable | BAL PD Response |
| Fixed continuous independent variable | Baseline*PD marker |
| Fixed categorical independent variables | Treatment*PD marker |

Information on the effects and prior distributions for parameters:

| Туре | Name (#Levels) | Parameters | Priors |
|---|---|---|---|
| Fixed | Baseline (2h) * | #1 Baseline (2h) * | N(Mean=0, Var=1E6) |
| Continuous | PD marker (2) | Ind[Total Protein = 1] | |
| | | #2 Baseline (2h) * | N(Mean=0, Var=1E6) |
| | | Ind[Neutrophil = 1] | |
| Fixed | Treatment * PD | #1 Placebo * | N(Mean=0, Var=1E6) |
| Categorical | marker (4) | Ind[Total Protein = 1] | |
| | | #2 Placebo * | N(Mean=0, Var=1E6) |
| | | Ind[Neutrophil = 1] | |
| | | #3 GSK2798745 * | N(Mean=0, Var=1E6) |
| | | Ind[Total Protein = 1] | |
| | | #4 GSK2798745 * | N(Mean=0, Var=1E6) |
| | | Ind[Neutrophil = 1] | |
| Random | Subjects | Separate value per | $\sigma_{Subject}^2$ ~Gamma(0.001,0.001) |
| | | subject, sampled as | |
| | | i.i.d. $\sim N(0, \sigma_{Subject}^2)$ | |

- The default prior for the VCV matrix would be an Inverse-Wishart with parameters k and S (where S = (k p 1) \* R and p = dimension of the VCV matrix). Under this framework, R can be thought of as a best guess for the VCV of the endpoints/timepoints being modelled. Care should be taken in the choice of k and R for each endpoint to ensure it is uninformative.
- Separate variance-covariance matrices will be used for treatment groups if there is sufficient

- information/data to allow for this (i.e. convergence occurs for all parameters and values do not get "stuck" at zero) to obtain separate estimates for the correlation between the endpoints. If there is not sufficient information then the default position is for treatment groups to share a common variance-covariance matrix.
- An optional exploration/model building step may take place by adding other covariates to the
  model that may explain a significant proportion of variance in the response and/or imbalance
  between treatment groups at baseline and/or be justified by biological rationale/expert
  judgment or statistical tools (raw plots and model selection criteria). Only the results of the final
  model would be reported in the Clinical Study Report (CSR).
- For the final model, appropriate combinations of model parameters should be combined to obtain treatment effects of interest, including performing any back-transformations that are required. For example, assuming log<sub>e</sub> transformation is required, the percentage change for GSK2798745 relative to placebo in 26h total protein will be obtained by computing exp(β<sub>GSK2798745,Total Protein</sub> β<sub>Placebo,Total Protein</sub>) for each MCMC iteration, which should be programmed between the BEGINNODATA and ENDNODATA statements (within PROC MCMC procedure).
- To obtain probability statements for parameters/effects of interest use binary flag variables. For
  each MCMC iteration if the condition is satisfied the iteration is flagged as a 1, if not it is
  flagged as 0. The proportion of iterations flagged as 1 gives the posterior probability of the
  statement of interest i.e. the proportion of MCMC iterations for which the percentage reduction
  in the BAL biomarker for GSK2798745 c.f. placebo for the specified sampling timepoint is
  greater than zero.
- For example, the SAS syntax for computing the flag for any percentage reduction in BAL total protein as well as neutrophils would be: flagsuccess\_TPROTNEU = (ratio\_TPRO < 1 and ratio\_TNEU < 1); . Where ratio\_TPRO is the parameter used to store the ratio of adjusted posterior medians for GSK2798745 relative to placebo for total protein, calculated as exp(β<sub>GSK2798745,Total Protein</sub> β<sub>Placebo,Total Protein</sub>) and flagsuccess\_TPROTNEU being the binary variable where any percentage reduction in both total protein and total neutrophil , active relative to placebo, flags success. This will be computed for a number of different effects of interest: 10%, 25% percentage reduction, etc

#### **Model Checking & Diagnostics**

See Section 7.1.5.1 (Model Checking and Diagnostics)

#### Model Results Presentation

- Point estimates (median values of posterior distributions), the standard deviation of the
  posterior distribution (SDs) and 95% credible intervals (CrI) intervals will be presented for each
  treatment group and treatment comparison (absolute and percentage change) at each
  sampling time point. A number of posterior probability statements will also be expressed, as
  described in Table 2 of Section 7.2.5.1 (Model Results Presentation) for each timepoint.
- Point estimates for each treatment group and treatment comparison (absolute and percentage change) for each endpoint will be expressed graphically. See Appendix 11: List of Data Displays for example displays.
- The joint posterior probability statements of interests in Table 2 were correct at the time of writing but may not be limited to these listed.

| Posterior Probability Statement (where | Interpretation |
|---|---|
| X <sub>TP</sub> = treatment ratio of GSK2798745 / | morprotation |
| Pbo for 26h total protein) | |
| PP ( $X_{TP} \le 0.25$ and $X_{NE} \le 0.25$ ) | Posterior probability of at least a 75% |
| 11 (MP = 0.20 and MP = 0.20) | reduction in both mean BAL total protein and |
| | total neutrophil counts for GSK2798745 |
| | relative to placebo |
| PP ( $X_{TP} \le 0.5 \text{ and } X_{NE} \le 0.5$ ) | Posterior probability of at least a 50% |
| 11 (ATP = 0.0 and ANE = 0.0) | reduction in both mean BAL total protein and |
| | total neutrophil counts for GSK2798745 |
| | relative to placebo |
| PP ( $X_{TP} \le 0.75$ and $X_{NE} \le 0.75$ ) | Posterior probability of at least a 25% |
| ( = 0 0 0 0 7445 = 0 0) | reduction in both mean BAL total protein and |
| | total neutrophil counts for GSK2798745 |
| | relative to placebo |
| PP ( $X_{TP} \le 0.9$ and $X_{NE} \le 0.9$ ) | Posterior probability of at least a 10% |
| ( the one show that | reduction in both mean BAL total protein and |
| | total neutrophil counts for GSK2798745 |
| | relative to placebo |
| $PP(X_{TP} \le 1 \text{ and } X_{NE} \le 1)$ | Posterior probability of any reduction in both |
| ( ) | mean BAL total protein and total neutrophil |
| | counts for GSK2798745 relative to placebo |
| PP ( $X_{TP} > 1$ and $X_{NE} > 1$ ) | Posterior probability of any increase in both |
| , | mean BAL total protein and total neutrophil |
| | counts for GSK2798745 relative to placebo |
| PP ( $X_{TP} > 1.1 \text{ and } X_{NE} > 1.1$ ) | Posterior probability of at least a 10% increase |
| | in both mean BAL total protein and total |
| | neutrophil counts for GSK2798745 relative to |
| | placebo |
| PP ( $X_{TP} > 1.25$ and $X_{NE} > 1.25$ ) | Posterior probability of at least a 25% increase |
| , | in both mean BAL total protein and total |
| | neutrophil counts for GSK2798745 relative to |
| | placebo |
| PP ( $X_{TP} > 1.5$ and $X_{NE} > 1.5$ ) | Posterior probability of at least a 50% increase |
| | in both mean BAL total protein and total |
| | neutrophil counts for GSK2798745 relative to |
| | placebo |
| PP ( $X_{TP} > 1.75$ and $X_{NE} > 1.75$ ) | Posterior probability of at least a 75% increase |
| | in both mean BAL total protein and total |
| | neutrophil counts for GSK2798745 relative to |

• **PD\_F2**: The correlation between endpoints for each treatment arm will be extracted from the statistical analysis and displayed on a panel scatter plot showing 26h total protein against 26h total neutrophils, with separate panels for treatment arm (as it is anticipated the relationship between endpoints will be different between treatment arms).

### 8. SAFETY ANALYSES

The safety analyses will be based on the All Subjects population, unless otherwise specified.

## 8.1. Adverse Events Analyses

Adverse events analyses including the analysis of adverse events (AEs), Serious (SAEs) and other significant AEs will be based on GSK Core Data Standards. The details of the planned displays are provided in Appendix 11: List of Data Displays.

# 8.2. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of Chemistry laboratory tests, Hematology laboratory tests, Urinalysis, and liver function tests will be based on GSK Core Data Standards. The details of the planned displays are in Appendix 11: List of Data Displays.

# 8.3. Other Safety Analyses

The analyses of non-laboratory safety test results including ECGs and vital signs will be based on GSK Core Data Standards, unless otherwise specified.

The CSSRS questionnaire will be summarised using a listing and summary table. FOBT results will summarised using a listing and summary table.

The details of the planned displays are presented in Appendix 11: List of Data Displays

#### 9. PHARMACOKINETIC ANALYSES

# 9.1. Primary Pharmacokinetic Analyses

#### 9.1.1. Endpoint / Variables

#### 9.1.1.1. Drug Concentration Measures

Refer to Appendix 5: Data Display Standards & Handling Conventions (Section 12.5.3 Reporting Standards for Pharmacokinetic)

#### 9.1.1.2. Derived Pharmacokinetic Parameters

Pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices and using the currently supported version of WinNonlin. All calculations of non-compartmental parameters will be based on actual sampling times. Pharmacokinetic parameters listed will be determined from the plasma concentration-time data, as data permits.

| Parameter | Parameter Description |
|-----------|-------------------------------------|
| Cmax | Plasma GSK2798745 for Day 1 |
| Tmax | Plasma GSK2798745 for Day 1 |
| AUC(0-26) | Plasma GSK2798745 for Day 1 & Day 2 |

#### NOTES:

• Additional parameters may be included as required.

## 9.1.2. Population of Interest

The primary pharmacokinetic analyses will be based on the pharmacokinetic population, unless otherwise specified.

### 9.1.3. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 11: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 9.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

# 9.2. Secondary Pharmacokinetic Analyses

### 9.2.1. Endpoint / Variables

#### 9.2.1.1. Drug Concentration Measures

Refer to Appendix 5: Data Display Standards & Handling Conventions (Section 12.5.3 Reporting Standards for Pharmacokinetic)

## 9.2.1.2. Derived Pharmacokinetic Parameters

Pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices and using the currently supported version of WinNonlin. All calculations of non-compartmental parameters will be based on actual sampling times. Pharmacokinetic parameters listed will be determined from the plasma concentration-time data, as data permits.

| Parameter | Parameter Description |
|-----------|----------------------------------------|
| Cmax | Plasma metabolite GSK3526876 Day 1 |
| Tmax | Plasma metabolite GSK3526876 Day 1 |
| AUC(0-26) | Plasma metabolite GSK3526876 Day 1 & 2 |
| BAL 2h | BAL metabolite GSK3526876 Day 1 |
| BAL 26h | BAL metabolite GSK3526876 Day 1 |
| BAL 2h | BAL GSK2798745 concentration at 2h |
| BAL 26h | BAL GSK2798745 concentration at 26h |

#### NOTES:

Additional parameters may be included as required.

## 9.2.2. Population of Interest

The secondary pharmacokinetic analyses will be based on the pharmacokinetic population, unless otherwise specified.
# 10. PHARMACOKINETIC / PHARMACODYNAMIC ANALYSES

The primary goal of this analysis is to characterize the pharmacokinetic / pharmacodynamic relationship of GSK2798745 administered orally in the participants.

# 10.1. Statistical Analyses / Methods

A summary of the planned pharmacokinetic / pharmacodynamic analyses are outlined below:

- Individual plasma GSK2798745 Cmax, will be plotted against corresponding BAL 2h GSK2798745 drug levels. Analysis may be undertaken to assess relationship of drug levels in plasma and target site (BAL).
- Individual plasma GSK2798745 AUC(0-26) and C26 data will be plotted against BAL 26h GSK2798745 drug levels. Regression analysis will be undertaken to assess relationship of drug levels in plasma and target site (BAL)
- Individual plasma GSK2798745 AUC(0-26), C26 and C<sub>max</sub> data will be plotted against total BAL protein at 26h (primary clinical endpoint). Placebo treatment data (i.e. 0 drug concentration and corresponding total BAL protein will also be included in the PK-PD analysis. Analysis may be undertaken to evaluate the association between GSK2798745 PK parameters and change in BAL total protein.

Data specifications for PK/PD analyses presented in Appendix 11: Pharmacokinetic / Pharmacodynamic Analyses.

# 11. REFERENCES

Costa M, Fortunato L, Abellan J, Chen G, He Z, Archer G. Bayesian Statistics Best Practice at GSK – Clinical Trials using Bayesian Inference. GlaxoSmithKline; 2017.

Holz O, Tan L, Schaumann L, Müller M, Scholl D, Hidi R, et al. Inter- and intrasubject variability of the inflammatory response to segmental endotoxin challenge in healthy volunteers. *Pulmonary Pharmacology & Therapeutics*. 2015;35:50-9.

# 12. APPENDICES

# 12.1. Appendix 1: Protocol Deviation Management and Definitions for Evaluable Population

# 12.1.1. Exclusions from Evaluable Population

Subjects with major/important protocol deviations will be excluded from Evaluable Population. The Protocol Deviation Management Plan (PDMP) will be used to determine major/important protocol deviations that will lead to exclusion from the Evaluable Population.

# 12.2. Appendix 2: Schedule of Activities

#### 12.2.1. Protocol Defined Schedule of Events

- The timing and number of planned study assessments, including safety, pharmacokinetic, pharmacodynamics and exploratory biomarker assessments may be altered during the course of the study based on newly available data (e.g., to obtain data closer to the time of peak plasma concentrations) to ensure appropriate monitoring.
- Any changes in the timing or addition of time points for any planned study assessments must be documented and approved by the relevant study team member and then archived in the sponsor and site study files, but will not constitute a protocol amendment. The IRB/IEC will be informed of any safety issues that require alteration of the safety monitoring scheme or amendment of the informed consent form (ICF).

# 12.2.2. Screening

| | Screening<br>(Days –28 to –2) |
|-------------------------------------|-------------------------------|
| Outpatient visit | X |
| Informed consent | X |
| Inclusion and exclusion criteria | X |
| Demography | X |
| Full physical examination | X |
| Height and weight | X |
| Medical history | X |
| Past and current medical conditions | X |
| HIV, Hepatitis B and C screening | X |
| FSH and oestradiol <sup>1</sup> | X |
| Drug, alcohol and cotinine screen | X |
| C-SSRS | X |
| Laboratory assessments <sup>2</sup> | X |
| 12-lead ECG <sup>3</sup> | X |
| Vital signs <sup>4</sup> | X |
| Spirometry <sup>5</sup> | X |
| FOBT <sup>6</sup> | X |

C-SSRS: Columbia Suicide Severity Rating Scale; ECG: electrocardiogram; FOBT: Faecal Occult Blood Test; HIV: human immunodeficiency virus.

- 1. Postmenopausal females whose postmenopausal status is in doubt only.
- 2. Haematology, clinical chemistry (including liver chemistry), cardiac troponins, urinalysis and coagulation profile.
- 3. In triplicate.
- 4. Blood pressure and heart rate in triplicate. Single temperature measurement.
- 5. Forced expiratory volume in 1 second (FEV1) and forced vital capacity (FVC). Triplicate measurement, the highest of which should be recorded in the case report form.
- 6. May be measured during the screening window or on Day –1. FOBT cards will be provided at screening and must be returned to the laboratory and analysed before dosing.

# 12.2.3. Treatment period

| | Day –1 <sup>2</sup> | | | | | Day 1 | 1 | | | | | Day 2 <sup>1</sup> | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Pre-<br>dose | 0 h | 1 h | 2 h | 3 h | 6 h | 8 h | 12 h | 14 h | 25.5 h | 26 h | 30 h | Day 4 |
| Inpatient stay <sup>2</sup> | | ←=== | ===== | ===== | ===== | ===== | ===== | ===== | ===== | ===== | ====== | ===== | ===→ | |
| Telephone call <sup>3</sup> | | | | | | | | | | | | | | X |
| Drug, alcohol and cotinine screen | Χ | | | | | | | | | | | | | |
| Laboratory assessments <sup>4</sup> | Х | | | | | | | | | | | | Χ | |
| 12-lead ECG <sup>5</sup> | Χ | Χ | | | | | | | | | | | Χ | |
| Blood pressure and heart rate <sup>5</sup> | Χ | Χ | | Х | | | Х | | Х | Χ | | | Χ | |
| Temperature <sup>6</sup> | X | Χ | | Х | Χ | | Х | Χ | X | Χ | | | Χ | |
| Spirometry <sup>7</sup> | Χ | Χ | | | | | Х | | | | Х | | Χ | |
| C-SSRS | | | | | | | | | | | | | Χ | |
| Randomisation | | Χ | | | | | | | | | | | | |
| Study treatment | | | Х | | | | | | Х | | | | | |
| Pulse oximetry <sup>8</sup> | | | | | Х | | | | | | | Χ | | |
| Bronchoscopy, baseline BAL and challenge <sup>9</sup> | | | | | X | | | | | | | | | |
| Bronchoscopy and post-challenge BAL <sup>10</sup> | | | | | | | | | | | | Х | | |
| Blood sample for exploratory biomarkers <sup>11</sup> | | | | | X <sup>11</sup> | Х | | Х | | | | X <sup>11</sup> | | |
| Blood sample for PK | | | | | | S | ee foo | tnote 12 | | | | | | |
| AE review | | <b>←===</b> | ===== | ==== | ===== | ==== | ===== | | | ===== | ====== | | ====== | ==== |
| SAE review | ←===== | ====== | ===== | | ===== | | ===== | | | | ====== | ===== | | ==== |
| Concomitant medication review | ←===== | ====== | ===== | | ===== | | ===== | | | | ====== | ====== | | ==== |

AE: adverse event; BAL: bronchoalveolar lavage; ECG: electrocardiogram; PK: pharmacokinetic; SAE: serious adverse event, C-SSRS: Columbia Suicide Severity Rating Scale.

- 1. Time points relative to the first dose on Day 1.
- 2. Admission on Day –1, at a time to allow all Day –1 procedures to be done; discharge on Day 2, at least 4 h after the bronchoscopy.
- 3. To check for any AEs.
- 4. Haematology, clinical chemistry (including liver chemistry), cardiac troponins, urinalysis and coagulation profile.
- 5. Triplicate on Day-1 and pre-dose. Single measurements at time points after dosing.
- 6. Immediately before BAL sampling/LPS challenge at the 2-h time point.
- 7. Forced expiratory volume in 1 second (FEV1) and forced vital capacity (FVC). Triplicate measurements at each time point, the highest of which should be recorded in the case report form.
- 8. Pulse oximetry to be measured during bronchoscopy procedures. Only AEs to be recorded.
- 9. BAL samples for total protein, neutrophil counts, GSK2798745 and exploratory biomarkers. Baseline BAL sample from a segment in the left lower lobe, followed by segmental challenge of the lungs: LPS in right middle segment; saline control in the lingula segment of the contralateral side. Challenges to be done as close as possible to 2 h post-dose.
- 10. BAL samples for total protein, neutrophil counts, GSK2798745 and exploratory biomarkers. Baseline and post-dose measurements to be done by the same person, where possible.
- 11. Blood samples for exploratory biomarkers. The 2- and 26-h blood samples should be taken immediately before BAL sampling.
- 12. PK samples will be taken pre-dose and at 0.5, 1, 1.5, 2, 2.5, 3, 6, 8, 12, 12.5, 13, 13.5, 14, 15, 24 and 26 h after the first dose. The 2- and 26-h blood sample should be taken immediately before BAL sampling

# 12.2.4. Follow-up/Early Withdrawal

| | Follow-up/Early Withdrawal (Day 8 [± 1 day]) |
|---|---|
| Outpatient visit | X |
| Full physical examination | Х |
| Weight | X |
| Laboratory assessments <sup>1</sup> | X |
| 12-lead ECG <sup>2</sup> | X |
| Vital signs <sup>3</sup> | X |
| Spirometry <sup>4</sup> | X |
| FOBT <sup>5</sup> | X |
| AE review | X |
| SAE review | X |
| Concomitant medication review | X |

AE: adverse event; ECG: electrocardiogram; FOBT: Faecal Occult Blood Test; SAE: serious adverse event.

- 1. Haematology, clinical chemistry (including liver chemistry), cardiac troponins and urinalysis.
- 2. Single measurement.
- 3. Blood pressure, heart rate, temperature. Single measurement.
- 4. Forced expiratory volume in 1 second (FEV1) and forced vital capacity (FVC). Triplicate measurement, the highest of which should be recorded in the case report form.
- 5. FOBT cards will be provided upon discharge from the unit and should be returned by the follow-up/early withdrawal visit.

# 12.3. Appendix 3: Assessment Windows

# 12.3.1. Definitions of Assessment Windows for Analyses

Refer to the Study Reference Manual (SRM) for acceptable time deviation windows for study assessments and procedures.

26h PK blood samples that are taken outside of 25.5h-26.5h will be excluded from plasma concentration by time point summary tables as well as displays that include planned timepoint. The 26h blood PK sample has a wider acceptable time deviation window than other blood PK samples due to the requirement for the sample to be aligned with the 26h BAL sample. This may impact on PK summaries.

# 12.4. Appendix 4: Study Phases and Treatment Emergent Adverse Events

# 12.4.1. Study Phases

Assessments and events will be classified according to the time of occurrence relative to the two study treatment doses and LPS/saline challenges.

| Study Phase | Definition |
|----------------|---------------------------------------------|
| Pre-Treatment | Date/Time ≤ Study Treatment Start Date/Time |
| Post-Treatment | Study Treatment Start Date/Time < Date/Time |

#### NOTES:

Study Treatment Start relates to the 1st dose received by the individual.

#### 12.4.1.1. Study Phases for Concomitant Medication

| Study Phase | Definition |
|---|---|
| Prior | If medication end date is not missing and is before 28 days prior to screening visit |
| Concomitant | Any medication that is not a prior |

#### NOTES:

• Please refer to Appendix 7: Reporting Standards for Missing Data for handling of missing and partial dates for concomitant medication. Use the rules in this table if concomitant medication date is completely missing.

# 12.4.2. Treatment and LPS Emergent Flag for Adverse Events

The flag assigned to a participant's AE will depend upon the type of AE, the magnitude of the AE and the study phase the AE occurred in. Each adverse event will be considered on a case-by-case basis.

# 12.5. Appendix 5: Data Display Standards & Handling Conventions

#### 12.5.1. Reporting Process

| Software | Software |
|---|---|
| The currently supply | orted versions of SAS software and R will be used. |
| Reporting Area | Reporting Area |
| HARP Server | : UK1SALX00175.corpnet2.com |
| HARP Compound | : \ARPROD\GSK2798745\207464\Internal_01 : \ARPROD\GSK2798745\207464\Internal_02 : \ARPROD\GSK2798745\207464\Headline : \ARPROD\ GSK2798745\207464\Final |
| Analysis Datasets | |

# Analysis datasets will be created according to legacy GSK A&R dataset standards.

statistical analyses results easier.

- Intermediate Datasets
   The following instructions are recommended to make modelling and tracking of
- The Bayesian framework necessitates the storage of intermediate outputs datasets
   (convention dictates that they be stored in the dddata folder of the reporting effort). It
   is strongly recommended that a file naming convention be adopted across all
   MCMC analyses to allow easy grouping/location of associated items. The naming
   convention has to follow the SAS dataset length rules, and any HARP naming
   conventions.
- The file name is made up of components joined by underscores. This should allow items to automatically group/sort when viewed as a list.
- The components of the file name may change and is included for guidance.

| Component ID | Description | Examples | Clarification |
|---|---|---|---|
| 1 | Three letters for the sample matrix | BAL<br>BLD | Bronchoalveolar Lavage Blood |
| 2 | Item/Analyte | TPRO TNEU DNEU TALB <bicat code=""></bicat> | Total Protein Total Neutrophil Count Differential Neutrophil Count Total Albumin Count <taken dataset="" from="" si=""></taken> |
| 3 | Single digit Population code | 1<br>2<br>etc | All Subjects Evaluable (Statistician will need to track assignments) |

| Component ID | Description | Examples | Clarification |
|---|---|---|---|
| 4 | Single digit Model ID | 1 | Primary Analysis |
| | (may vary depending on the | 2 | Sensitivity Analysis 1 |
| | analysis, so model 1 can | etc | (Statistician will need to track |
| | have different meanings | | assignments on a per |
| | across objectives/sample | | objectives/sample |
| | matrices/endpoints) | | matrices/endpoint basis) |
| 5 | Double digit Analysis ID | 01 | Statistician will need to track |
| | (specific to the model) | 02 | on a per item basis |
| | | 03 | |
| | | 04 | |
| | | etc | |
| 6 | MCMC related item | poall | Posterior Summary Stats (processed and ready for display) |
| | | pokdein | Posterior samples |
| | | + Others as required | |

 Example for the output dataset produced from PROC MCMC with summary statistics used for T/L/F for the Primary analysis of 26h BAL Total Protein using the Evaluable population using the simplest model (only intercept, baseline and treatment group as covariates): "BAL TPRO 3 1 01 poall"

#### **Generation of RTF Files**

RTF files will be generated for the final reporting effort.

# 12.5.2. Reporting Standards

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location: https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics
- Do not include participant level listings in the main body of the GSK Clinical Study Report. All
  participant level listings should be located in the modular appendices as ICH or non-ICH listings

#### **Formats**

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and

- calculation of any derived parameters, unless otherwise stated.
- The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the participant's listings.

#### **Unscheduled Visits**

- Unscheduled visits will not be included in summary tables and/or figures.
- All unscheduled visits will be included in listings.

# Descriptive Summary Statistics Continuous Data Refer to IDSL Statistical Principle 6.06.1 Categorical Data N, n, frequency, %

#### **Graphical Displays**

- Refer to IDSL Statistical Principles 7.01 to 7.13.
- Where appropriate, specific SAS attribute maps and formats should be applied to treatments groups or subjects to allow standardisation of graphics. Specific subject level attributes allow tracking and distinguishing subjects across displays and aids interpretation.
- Please consult with GSK statistician to obtain final attributes map.
- Treatment attributes:

| Treatment | Colour | Plotting Symbol | Line Style |
|------------|--------|----------------------|------------|
| Placebo | Blue | Circle, Solid | Solid |
| GSK2798745 | Red | Triangle (up), Solid | Solid |

Example of subject attributes:

| Subject | Colour | Plotting Symbol | Line Style |
|---------|--------|------------------|------------|
| PPD | Cyan | Diamond (filled) | Solid |
| | Salmon | Asterisk | Dashed |

# 12.5.3. Reporting Standards for Pharmacokinetic

| Pharmacokinetic Con | Pharmacokinetic Concentration Data |
|---|---|
| PC Windows Non-<br>Linear (WNL) File | PC WNL file (CSV format) for the non compartmental analysis by Clinical Pharmacology Modelling and Simulation function will be created according to GUI_51487. Note: Concentration values will be imputed as per GUI_51487 |
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | Refer to IDSL PK Display Standards. Refer to IDSL Statistical Principle 6.06.1. Note: Concentration values will be imputed as per GUI_51487 for descriptive summary statistics/analysis and summarized graphical displays only. |
| NONMEM/Pop PK<br>File | Not applicable. |
| Pharmacokinetic Para | ameter Derivation |
| PK parameters to be provided to programmer | The following PK parameters will be derived by CPMS and provided to the programmer: [PK parameters, as defined in Section 9.1.1.2 and Section 9.2.1.2)] |

| Pharmacokinetic Para | Pharmacokinetic Parameter Data |
|---|---|
| Is NQ impacted PK<br>Parameters Rule<br>Being Followed | Yes, refer to Standards for Handling NQ Impacted PK Parameters, December 2009. |
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | Refer to IDSL PK Display Standards. |

#### 12.6. Appendix 6: Derived and Transformed Data

#### 12.6.1. General

#### **Multiple Measurements at One Analysis Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- If there are two values within a time window (as per Section 12.3.1) the value closest to the target day for that window will be used. If values are the same distance from the target, then the mean will be taken.
- Participants having both High and Low values for Normal Ranges at any post-baseline visit for safety parameters will be counted in both the High and Low categories of "Any visit post-baseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

#### Study Day

- Calculated as the number of days from First Dose Date:
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < First Dose Date → Study Day = Ref Date First Dose Date
  - Ref Data ≥ First Dose Date → Study Day = Ref Date (First Dose Date) + 1

#### 12.6.2. Study Population

#### **Treatment Compliance**

Treatment compliance is defined as a participant receiving both doses of study treatment (0 h and 12 h).

# Challenge Compliance

 Challenge compliance is defined as undergoing segmental challenge to the lungs, via bronchoscopy, at 2 hours after the first dose of investigational medicinal product (IMP): 10 mL LPS (4 ng/kg) instilled into the right middle segment and 10 mL saline control instilled into the lingula segment of the contralateral side.

# 12.6.3. Pharmacodynamic and Biomarker

#### **Derivation of BAL White Blood Cell Counts and Differentials**

 Differential cell count gives the relative percentage of each type of white blood cell and is calculated as follows.

 $Differential\ cell\ type\ count\ (\%) = \frac{Total\ cell\ type\ count\ (cells/mL)}{Total\ white\ blood\ cell\ (leukocyte)\ count\ (cells/mL)}$ 

Equivalently, to calculate absolute cell type count:

#### **Derivation of BAL White Blood Cell Counts and Differentials**

Total cell type count (cells/mL) = Differential cell type count (%)  $\times$  total WBC count (cells/mL)

- It is anticipated that pharmacodynamic endpoints and biomarkers will require log-transformation in all analyses to improve model fitting. Following model fitting, back-transformation will occur and treatment effects (GSK2798745 relative to placebo) will be expressed as percentage changes.
- Percentage change, active relative to placebo, will be calculated as:

$$Percentage change = \left(\frac{Active \ adjusted \ posterior \ median}{Placebo \ adjusted \ posterior \ median} - 1\right) \times 100$$

Ratio, active relative to placebo, will be calculated as:

• Urea concentration data in plasma and BAL will be used to calculate the dilution effect of the lavage which is used to extract the sample from the lung compartment. A correction for dilution will be applied to all BAL analytes to derive corrected concentrations i.e. each BAL analyte will be adjusted to account for the magnitude of dilution during the BAL procedure using urea plasma concentration as a reference point. A dilution factor for each BAL sample will be calculated as BAL urea concentration / plasma urea concentration. Each BAL analyte will be multiplied by this dilution factor to "correct". Outputs for BAL analytes adjusted for dilution factor may be produced as an exploratory analysis (See Appendix 11: List of Data Displays). Corrected BAL concentrations for dilution factor will be derived as follows:

Corrected concentration (pg/ml) = BAL concentration  $(pg/ml) \times Dilution$  factor

Where,

Dilution factor = 
$$\frac{Urea\ plasma\ concentration}{Urea\ BAL\ concentration}\ at\ time\ (t)$$

# 12.7. Appendix 7: Reporting Standards for Missing Data

# 12.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Participant study completion (i.e. as specified in the protocol) was defined as completing all phases of the study including the follow-up visit.</li> <li>Withdrawn participants may be replaced in the study.</li> </ul> |
| | All available data from participants who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified. |
| | Withdrawal visits will be slotted as per Appendix 3: Assessment Windows or will be summarised as withdrawal visits. |

# 12.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: |
| Outliers | Any participants excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |
| BAL<br>Pharmacodynamic<br>endpoints | No missing data will be imputed. |
| Blood<br>Pharmacodynamic<br>endpoints | <ul> <li>Responses unquantifiable due to being below LLQ will be imputed as ½ LLQ.</li> <li>Responses above ULQ will be imputed as ULQ.</li> </ul> |

# 12.7.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in participant listing displays. |
| Concomitant<br>Medications/<br>Medical<br>History | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> </li> <li>The recorded partial date will be displayed in listings.</li> </ul> |

#### 12.7.2.2. Handling of Missing Data for Statistical Analysis

For BAL endpoints, any participant that has missing data for baseline (2h) or 26h (LPS lobe) does not meet the criteria to be included in the evaluable population and therefore will be excluded from the analysis. No imputation will be performed.

For analyses of repeated measures data (blood biomarkers), responses that are unquantifiable due to being below LLQ will be imputed as ½ LLQ and above ULQ will be imputed as ULQ, whilst for any other missing data SAS PROC MCMC automatically assumes/implements a missing at random/multiple imputation approach if any of the supplied response variables are missing. Given this is a proof of mechanism study, this is deemed sufficient.

# 12.8. Appendix 8: Values of Potential Clinical Importance

# 12.8.1. Laboratory Values

| Hematology | | | |
|---|---|---|---|
| Analyte | Effect | Relative – Low<br>(Multipliers of LLN) | Relative – High<br>(Multipliers of ULN) |
| White Blood Cell Count (x109/ L) | | 0.67 | 1.82 |
| Neutrophil Count (x10 <sup>9</sup> / L) | | 0.83 | |
| | Male | | 1.03 |
| Hemoglobin (g/L) | Female | | 1.13 |
| Hamatacrit (ratio of 1) | Male | | 1.02 |
| Hematocrit (ratio of 1) | Female | | 1.17 |
| Platelet Count (x109/ L) | | 0.67 | 1.57 |
| Lymphocytes (x10 <sup>9</sup> / L) | | 0.81 | |
| Monocytes (x10 <sup>9</sup> / L) | | 0.5 | 1.8 |
| Red Blood Cell Count (x109/ L) | | 0.7 | 1.7 |
| Reticulocytes (%) | | 0 | 1.5 |

| Chemistry | | | |
|---|---|---|---|
| Analyte | Effect | Relative – Low<br>(Multipliers of LLN) | Relative – High<br>(Multipliers of ULN) |
| Calcium (mmol/L) | | 0.91 | 1.06 |
| Glucose (mmol/L) | | 0.71 | 1.41 |
| Potassium (mmol/L) | | 0.86 | 1.10 |
| Sodium (mmol/L) | | 0.96 | 1.03 |
| Blood Urea Nitrogen (mmol/L) | | 0.7 | 1.5 |
| Total Protein (mg/dL) | | 0.6 | 1.7 |
| Creatinine phosphokinase (IU/L) | | 0 | 1.8 |
| Direct Bilirubin (umol/L) | | 0 | 1.6 |
| Analyte | Effect | Relative – Low<br>(Absolute Value) | Relative – High<br>(Absolute Value) |
| Creatinine (umol/L) | Chg from Baseline | | > 44 umol/L |

# **Urinalysis:**

During the study, a dipstick result (positive or negative) will be recorded for each participant at each timepoint. If the dipstick result is positive, a microscopy will be performed. The urinalysis dipstick result at day 8 and day 2 will be compared with day -

1 (pre-dose) and data of PCI will be flagged where a result changes from negative to positive and/or a microscopy is performed.

#### **Faecal Occult Blood Test:**

FOBT is performed at screening and follow-up with measurement as haemoglobin (iFOBT) ng/ml. Any positive haemoglobin measurement ( $\geq$ 50ng/ml) will be flagged as potentially clinically important and all results for a participant with at least one flagged result will appear in listings.

| Liver Function | | | |
|--------------------|---------|----------|-------------------------|
| Test Analyte | Units | Category | Clinical Concern Range |
| ALT/SGPT | U/L | High | ≥ 2x ULN |
| AST/SGOT | U/L | High | ≥ 2x ULN |
| AlkPhos | U/L | High | ≥ 2x ULN |
| T Bilirubin | µmol/L | High | ≥ 1.5x ULN |
| | μmol/L, | | ≥ 1.5x ULN T.Billirubin |
| T. Bilirubin + ALT | U/L | High | + |
| | U/L | | ≥ 2x ULN ALT |

| Other | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Cardiac Troponin (cTn) | Cardiac Troponin (cTn) ng/ml | | | >ULN or 2x Baseline<br>Value |
| Coagulation Profile | | | | |
| International Normalisation Ratio (INR) | | | < 0.85 | > 1.15 |
| Prothrombin Time (PTT) | % | | < 70 | > 120 |
| Fibrogen | g/l | | < 1.7 | > 4.2 |

#### 12.8.2. ECG

| ECG Parameter | Units | Clinical Concern Range | |
|-----------------------|----------|------------------------|-------|
| | | Lower | Upper |
| Absolute | Absolute | | |
| Absolute QTc Interval | msec | | >500 |
| Absolute PR Interval | msec | <110 | >220 |
| Absolute QRS Interval | msec | <75 | >110 |
| Change from Baseline | | | |

| ECG Parameter | Units | Clinical Co | oncern Range |
|----------------------------|-------|-------------|--------------|
| | | Lower | Upper |
| Increase from Baseline QTc | msec | | >60 |

# 12.8.3. Vital Signs

| Vital Sign Parameter | Units | Clinical Concern Range | |
|--------------------------|-------|------------------------|-------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | <85 | >160 |
| Diastolic Blood Pressure | mmHg | <45 | > 90 |
| Heart Rate | bpm | <50 | >110 |

| Vital Sign Parameter | Units | Clinical Concern Range | | | |
|---|---|---|---|---|---|
| (Change from Baseline) | | Decrease | | Increase | |
| | | Lower | Upper | Lower | Upper |
| Systolic Blood Pressure | mmHg | ≥20 | ≥40 | ≥20 | ≥40 |
| Diastolic Blood Pressure | mmHg | ≥10 | ≥20 | ≥10 | ≥20 |
| Heart Rate | bpm | ≥15 | ≥30 | ≥15 | ≥30 |

# 12.9. Appendix 9: Pharmacokinetic / Pharmacodynamic Analyses

# 12.9.1. Pharmacokinetic / Pharmacodynamic Dataset Specification

# Specification for PK-PD dataset [Proposed dataset name PKPD]

| Variable short name | Assessment description | Format | Unit | Valid Values / Format |
|---|---|---|---|---|
| С | Data Identifier | Integer | - | 0 |
| ID | Unique subject number | Numeric | | Different ID for different subject |
| STUD | Protocol Number | Integer | - | 207464 |
| SUBJ | Subject identifier in study | Integer | - | Maximum 10 characters (numeric or text). Different identifier for each subject |
| CENT | Study centre identifier | Integer | - | |
| DAY | Day of sampling | Integer | See<br>footnotes | See footnotes |
| C2 | Conc of<br>GSK2798745 2 h<br>post first dose | Decimal 3 d.p | ng/mL | Numeric – For placebo TRT arm C2 = 0 |
| C26 | Conc of<br>GSK2798745 26 h<br>post first dose | Decimal<br>3 d.p | ng/mL | Numeric - For placebo TRT arm C26 = 0 |
| AUC26 | Area under curve | Decimal | ng.h/mL | Numeric - For placebo TRT arm |
| | (0-26h) | 3 d.p | | AUC26 = 0 |
| Analyte | Drug analysed | Integer | - | GSK2798745 |
| Base_PD | Baseline corrected<br>BAL total protein<br>(i.e. before LPS<br>challenge and 2h<br>post dose | Decimal 3 d.p | - | BAL total protein |
| 745_PD | Corrected BAL total<br>protein at 26h post<br>dosing with<br>GSK2798745 (i.e.<br>24h post LPS<br>challenge) | Decimal 3 d.p | | BAL total protein |
| AGE | Age | Decimal | Yrs | Integer. Age in years at time of screening rounded down to give age at last birthday. |
| WT | Weight | Decimal | Kg | Weight in kilograms at time of screening. |
| BMI | Body mass index | Decimal | kg/m^2 | Body mass index calculated as weight divided by height squared |
| SEX | Subject gender | Integer | - | Integer. One of the following - 1 = Male |

| Variable short name | Assessment description | Format | Unit | Valid Values / Format |
|---|---|---|---|---|
| | | | | 2 = Female |
| SEXTEXT | Gender Identifier | Character | | M = Male, F=Female |
| TMT | Treatment identifier | Integer | - | Placebo = 0<br>GSK2798745 =1 |

# Data to be provided to CPMS as csv file shown below



C2: Conc of GSK2798745 2 h post dose

C26: Conc of GSK2798745 26 h post dose

AUC26: AUC(0-26h) GSK2798745

Base\_PD: Baseline corrected total BAL protein (i.e. before LPS challenge and 2h post dose

745\_PD: Corrected total BAL protein at 26h post dosing with GSK2798745 (i.e. 24h post LPS challenge)

# 12.10. Appendix 10: Abbreviations & Trade Marks

# 12.10.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| ALT/SGPT | Alanine Amino Transferase / Serum Glutamic-Pyruvic Transaminase |
| AST/SGOT | Aspartate Amino Transferase / Serum Glutamic Oxaloacetic |
| | Transaminase |
| A&R | Analysis and Reporting |
| BAL | Bronchoalveolar Lavage |
| BUN | Blood Urea Nitrogen |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| Crl | Credible Interval |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CRP | C-reactive Protein |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| CTR | Clinical Trial Register |
| CV <sub>b</sub> / CV <sub>w</sub> | Coefficient of Variation (Between) / Coefficient of Variation (Within) |
| DIC | Deviance Information Criterion |
| DBF | Database Freeze |
| DBR | Database Release |
| DOB | Date of Birth |
| DP | Decimal Places |
| eCRF | Electronic Case Record Form |
| EMA | European Medicines Agency |
| FDA | Food and Drug Administration |
| FDAAA | Food and Drug Administration Clinical Results Disclosure Requirements |
| GSK | GlaxoSmithKline |
| HPD | Highest Posterior Density |
| IA | Interim Analysis |
| ICH | International Conference on Harmonization |
| IDMC | Independent Data Monitoring Committee |
| IDSL | Integrated Data Standards Library |
| IL | Interleukin |
| IMMS | International Modules Management System |
| INR | International Normalisation Ratio |
| IP | Investigational Product |
| ITT | Intent-To-Treat |
| LLQ | Lower Limit of Quantification |
| LPS | Lipopolysaccharide |
| MCMC | Monte Carlo Markov Chain |
| MMRM | Mixed Model Repeated Measures |

| Abbreviation | Description |
|--------------|---------------------------------------------------|
| PCI | Potential Clinical Importance |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PK | Pharmacokinetic |
| PP | Per Protocol |
| PP | Posterior Probability |
| PopPK | Population PK |
| PTT | Prothrombin Time |
| QC | Quality Control |
| QTcF | Fridericia's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |
| RAMOS | Randomization & Medication Ordering System |
| SAC | Statistical Analysis Complete |
| SDSP | Study Data Standardization Plan |
| SDTM | Study Data Tabulation Model |
| SOP | Standard Operation Procedure |
| SP-B | Surfactant Protein B |
| TA | Therapeutic Area |
| TFL | Tables, Figures & Listings |
| TNF-alpha | Tumour Necrosis Factor alpha |
| ULQ | Upper Limit of Quantification |
| vWF | Von Willebrand Factor |

# 12.10.2. Trademarks

| Trademarks of the GlaxoSmithKline<br>Group of Companies |
|---------------------------------------------------------|
| HARP |
| RANDALL NG |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| NONMEM |
| R |
| SAS |
| WinNonlin |

# 12.11. Appendix 11: List of Data Displays

# 12.11.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|-----------------------------------|-------------|-------------|
| Study Population | 1.1 to 1.13 | |
| Pharmacodynamic and Biomarker | 2.1 to 2.17 | 2.1 to 2.29 |
| Safety | 3.1 to 3.18 | |
| Pharmacokinetic | 4.1 to 4.8 | 4.1 to 4.10 |
| Pharmacokinetic / Pharmacodynamic | | 7.1 to 7.2 |
| Section | List | tings |
| ICH Listings 1 to 32 | | |
| Other Listings | 33 | to 55 |

# 12.11.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required example mock-up displays provided in Appendix 12: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|-----------------------------------|---------|---------|----------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Pharmacodynamic and Biomarker | PD_Fn | PD_Tn | PD_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |
| Pharmacokinetic | PK_Fn | PK_Tn | PK_Ln |
| Pharmacokinetic / Pharmacodynamic | PKPD_Fn | PKPD_Tn | PK/PD_Ln |

#### NOTES:

• Non-Standard displays are indicated in the 'IDSL / Example Shell' or 'Programming Notes'.

#### 12.11.3. Deliverables

| | Delivery [Priority] [1] | Description |
|---|---|---|
| | IA1 [X] | Interim Analysis 1 |
| | IA2 [X] | Interim Analysis 2 |
| | HR [X] | Headline Results During Study (i.e. in-stream data review) |
| Ī | SAC [X] | Statistical Analysis Complete |

#### NOTES:

1. Indicates priority (i.e. order) in which displays will be generated for the reporting effort

# 12.11.4. Study Population Tables

| Study | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | |
| 1.1. | All Subjects | ES1 | Summary of Participant Disposition for the Participant Conclusion Record | ICH E3, FDAAA, EudraCT | SAC [1] |
| 1.2. | All Subjects | SD1 | Summary of Treatment Status and Reasons for Discontinuation of Study Treatment | ICH E3 | SAC [1] |
| 1.3. | Screened | ES6 | Summary of Screening Status and Reasons for Screen Failure | Journal Requirements | SAC [1] |
| Protoc | ol Deviation | | | | |
| 1.4. | All Subjects | DV1 | Summary of Important Protocol Deviations | ICH E3 | SAC [1] |
| Popula | ation Analysed | | | | |
| 1.5. | All Subjects | SP1 | Summary of Study Populations | IDSL | SAC [1] |
| 1.6. | All Subjects | SP2 | Summary of Exclusions from the Evaluable Population | IDSL | SAC [1] |
| Demog | graphic and Bas | eline Characteris | tics | | |
| 1.7. | All Subjects | DM1 | Summary of Demographic Characteristics | ICH E3, FDAAA, EudraCT | SAC [1] |
| 1.8. | All Subjects | DM11 | Summary of Age Ranges | EudraCT | SAC [1] |
| 1.9. | All Subjects | DM5 | Summary of Race and Racial Combinations | ICH E3, FDA, FDAAA, EudraCT | SAC [1] |
| Prior a | nd Concomitan | t Medications | | <b>'</b> | |
| 1.10. | All Subjects | MH1 | Summary of Past Medical Conditions | ICH E3 | SAC [1] |

| Study F | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.11. | All Subjects | MH1 | Summary of Current Medical Conditions | ICH E3 | SAC [1] |
| 1.12. | All Subjects | CM1 | Summary of Concomitant Medications | ICH E3 | SAC [1] |
| Exposu | Exposure and Treatment Compliance | | | | |
| 1.13. | FX1 ICH E3 | | | | |

# 12.11.5. Pharmacodynamic and Biomarker Tables

| Pharma | Pharmacodynamic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| BAL To | tal Protein | | | | |
| 2.1. | Evaluable | PD_T1 | Summary of <b>BAL Total Protein</b> by Timepoint (Baseline (2 h) and 26 h), Lung Lobe (LPS and Saline Challenge) and Treatment Group | Separate pages for arithmetic and geometric summary statistics. | IA1 [1], IA2 [1],<br>HR [1], SAC [1] |
| 2.2. | Evaluable | PD_T2 | 26 h BAL Total Protein: Summary of Posterior Distributions and Posterior Probability Statements from the Primary Analysis | Up to 4 pages. Page 1: Raw baseline values and baseline covariates values predictions are made at. Also add values used to determine predictions for any other covariates included in the model. Page 2: Adjusted posterior medians for each treatment group i.e. model adjusted predictions. 75% and 95% Crl. Page 3: Treatment comparisons in the form of adjusted posterior median absolute differences or percentage changes (dependent on endpoint and transformation). 75% and 95% Crl. Page 4: Posterior probability statements of interest. | IA [1], IA2 [1],<br>HR [1], SAC [1] |
| 2.3. | Evaluable | PD_T2 | Sensitivity Analysis: 26 h BAL Total Protein including 26 h Saline Lobe BAL Total Protein as a Covariate: Summary of Posterior Distributions and Posterior Probability Statements from the Primary Analysis | Conditional output. See programming notes above. | SAC [1] |

| Pharma | acodynamic: Ta | ables | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.4. | Evaluable | PD_T2 | Sensitivity Analysis: 26h BAL Total Protein Excluding Participants with High Saline Lobe BAL Total Protein Level: Summary of Posterior Distributions and Posterior Probability Statements from the Primary Analysis | Conditional output. See programming notes above. | SAC [1] |
| 2.5. | Evaluable | PD_T2 | 26 h BAL Total Protein and Total Neutrophil Count:<br>Summary of Posterior Distributions and Posterior Probability<br>Statements from the Multivariate Analysis | Conditional output. See programming notes above. | SAC [1] |
| BAL To | tal Neutrophil | Count | | | |
| 2.6. | Evaluable | PD_T1 | Summary of <b>BAL Total Neutrophil Count</b> by Timepoint (Baseline (2 h) and 26 h), Lung Lobe (LPS and Saline Challenge) and Treatment Group | Separate pages for arithmetic and geometric summary statistics. | HR [1], SAC [1] |
| 2.7. | Evaluable | PD_T2 | 26 h BAL Total Neutrophil Count: Summary of Posterior Distributions and Posterior Probability Statements from the Analysis | Up to 4 pages. Page 1: Raw baseline values and baseline covariates values predictions are made at. Also add values used to determine predictions for any other covariates included in the model. Page 2: Adjusted posterior medians for each treatment group i.e. model adjusted predictions. 75% and 95% Crl. Page 3: Treatment comparisons in the form of adjusted posterior median absolute differences or percentage changes (dependent on endpoint and transformation). 75% and 95% Crl. Page 4: Posterior probability statements of interest. | HR [1], SAC [1] |

| Pharma | Pharmacodynamic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| BAL Di | BAL Differential Neutrophil Count | | | | |
| 2.8. | Evaluable | PD_T1 | Summary of <b>BAL Differential Neutrophil Count</b> by Timepoint (Baseline (2 h) and 26 h), Lung Lobe (LPS and Saline Challenge) and Treatment Group | Separate pages for arithmetic and geometric summary statistics. | HR [1], SAC [1] |
| 2.9. | Evaluable | PD_T2 | 26h BAL Differential Neutrophil Count: Summary of Posterior Distributions and Posterior Probability Statements from the Analysis | Up to 4 pages. Page 1: Raw baseline values and baseline covariates values predictions are made at. Also add values used to determine predictions for any other covariates included in the model. Page 2: Adjusted posterior medians for each treatment group i.e. model adjusted predictions. 75% and 95% Crl. Page 3: Treatment comparisons in the form of adjusted posterior median absolute differences or percentage changes (dependent on endpoint and transformation). 75% and 95% Crl. Page 4: Posterior probability statements of interest. | HR [1], SAC [1] |
| Explora | atory BAL Biom | narkers | | | |
| 2.10. | Evaluable | PD_T1 | Summary of <b>Exploratory BAL Biomarkers (excluding WBCs)</b> by Timepoint (Baseline (2h) and 26h), Lung Lobe (LPS and Saline Challenge) and Treatment Group | One page per analyte. Separate pages for arithmetic and geometric summary statistics. | SAC [1] |

| Pharmacodynamic: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.11. | Evaluable | PD_T2 | 26h Exploratory BAL Biomarkers (excluding WBCs): Summary of Posterior Distributions and Posterior Probability Statements from the Analyses | Up to 4 pages per analyte. Page 1: Raw baseline values and baseline covariates values predictions are made at. Also add values used to determine predictions for any other covariates included in the model. Page 2: Adjusted posterior medians for each treatment group i.e. model adjusted predictions. 75% and 95% Crl. Page 3: Treatment comparisons in the form of adjusted posterior median absolute differences or percentage changes (dependent on endpoint and transformation). 75% and 95% Crl. Page 4: Posterior probability statements of interest. | SAC [1] |
| 2.12. | Evaluable | PD_T1 | Summary of BAL White Blood Cell Types (Totals and Differentials, except neutrophils): by Timepoint (Baseline (2h) and 26h), Lung Lobe (LPS and Saline Challenge) and Treatment Group | One page per analyte. Separate pages for arithmetic and geometric summary statistics. | SAC [1] |

| Pharma | acodynamic: Ta | ables | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.13. | Evaluable | PD_T2 | 26h BAL White Blood Cell Types (Totals and Differentials, except Neutrophils): Summary of Posterior Distributions and Posterior Probability Statements from the Analyses | Up to 4 pages per analyte. Page 1: Raw baseline values and baseline covariates values predictions are made at. Also. add values used to determine predictions for any other covariates included in the model. Page 2: Adjusted posterior medians for each treatment group i.e. model adjusted predictions. 75% and 95% Crl. Page 3: Treatment comparisons in the form of adjusted posterior median absolute differences or percentage changes (dependent on endpoint and transformation). 75% and 95% Crl. Page 4: Posterior probability statements of interest. | SAC [1] |
| BAL Ph | narmacodynam | ic/Biomarker Corr | ected for Dilution Factor | | |
| 2.14. | Evaluable | PD_T1 | Summary of All BAL Biomarkers Corrected for Dilution Factor by Timepoint (Baseline (2h) and 26h), Lung Lobe (LPS and Saline Challenge) and Treatment Group | Conditional output. One page per analyte. Separate pages for arithmetic and geometric summary statistics. | SAC [1] |
| 2.15. | Evaluable | PD_T2 | All BAL Biomarkers Corrected for Dilution Factor: Summary of Posterior Distributions and Posterior Probability Statements from the Analyses | Conditional output. See programming notes above. | SAC [1] |
| Explora | atory Blood Bio | markers | | | |
| 2.16. | Evaluable | PD_T1 | Summary of <b>Exploratory Blood Biomarkers</b> by Timepoint and Treatment Group | Separate pages for arithmetic and geometric summary statistics. | SAC [1] |

| Pharma | Pharmacodynamic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.17. | Evaluable | PD_T2 | Exploratory Blood Biomarkers: Summary of Posterior Distributions and Posterior Probability Statements from the Analyses | Approximately 7 pages per analyte. Add timepoint as first column. Page 1: Raw baseline values and baseline covariates values predictions are made at. Also. add values used to determine predictions for any other covariates included in the model. Page 2: Adjusted posterior medians at each timepoint i.e. model adjusted predictions. 75% and 95% Crl. Page 3: Treatment comparisons in the form of adjusted posterior median absolute differences or percentage changes (dependent on transformation) for each timepoint. 75% and 95% Crl. Page 4-7: Posterior probability statements of interest for '745 c.f. pbo – separate page for each timepoint. | SAC [1] |

# 12.11.6. Pharmacodynamic and Biomarker Figures

| Pharmaco | Pharmacodynamic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Populati<br>on | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| BAL Tota | l Protein | | | | |
| 2.1 | Evaluable | PD_F1 | <b>BAL Total Protein:</b> Geometric Means and 95% CI by timepoint and challenge (baseline, 26 h LPS Lobe, 26 h Saline Lobe) and treatment group | | IA [1], IA2 [1],<br>HR [1], SAC [1] |
| 2.2 | Evaluable | PD_F3 | <b>BAL Total Protein:</b> Participant Profiles of Baseline (2h) to 26h by Challenge and Treatment Group | Use participant attributes map so each subject has specific marker, line colour, pattern to track participant between plots. | IA [1], IA2 [1],<br>HR [1], SAC [1] |
| 2.3 | Evaluable | PD_F4 | <b>BAL Total Protein:</b> Point Estimates and Credible Intervals from the Primary Analysis | Separate pages for 75% and 95% Crl. Page to include 3 column panels. 1st: (Back-transformed) treatment group predictions, 2nd: Treatment group differences, 3rd: Percentage reduction ('745 c.f. Pbo). | IA [1], IA2 [1],<br>HR [1], SAC [1] |
| 2.4 | Evaluable | PD_F5 | <b>BAL Total Protein:</b> Posterior Distribution Density Plots from the Primary Analysis | 3 pages in total. Page 1: posteriors for separate treatment groups <b>overlaid</b> . Page 2: posterior for absolute difference (GSK2798745 c.f. placebo) Page 3: posterior for percentage reduction (GSK2798745 c.f. placebo) | IA [1], IA2 [1],<br>HR [1], SAC [1] |
| 2.5 | Evaluable | PD_F2 | Scatter plot of BAL 26h Total Protein v 26h Total Neutrophil counts | Overlay correlation coefficient from multivariate analysis (if performed) for each treatment group. | SAC [1] |

| Pharmace | Pharmacodynamic: Figures | | | | | | |
|---|---|---|---|---|---|--|--|
| No. | Populati<br>on | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] | | |
| BAL Tota | BAL Total Neutrophil Count | | | | | | |
| 2.6 | Evaluable | PD_F1 | <b>BAL Total Neutrophil Count:</b> Geometric Means and 95% CI by timepoint and challenge (baseline, 26 h LPS Lobe, 26 h Saline Lobe) and treatment group. | | HR [1], SAC [1] | | |
| 2.7 | Evaluable | PD_F3 | BAL Total Neutrophil Count: Participant Profiles of Baseline (2h) to 26h by Challenge and Treatment Group | Use participant attributes map so each subject has specific marker, line colour, pattern to track participant between plots. | HR [1], SAC [1] | | |
| 2.8 | Evaluable | PD_F4 | <b>BAL Total Neutrophil Count:</b> Point Estimates and 95% Credible Intervals from the Analysis | Page to include 3 column panels. 1st: (Back-transformed) treatment group predictions, 2nd: Treatment group differences, 3rd: Percentage reduction ('745 c.f. Pbo). | HR [1], SAC [1] | | |
| 2.9 | Evaluable | PD_F5 | BAL Total Neutrophil Count: Posterior Distribution Density Plots from the Analysis | 3 pages in total. Page 1: posteriors for separate treatment groups. Page 2: posterior for absolute difference (GSK2798745 c.f. placebo) Page 3: posterior for percentage reduction (GSK2798745 c.f. placebo) | HR [1], SAC [1] | | |
| BAL Diffe | rential Neutr | ophil Count | | | | | |
| 2.10 | Evaluable | PD_F1 | BAL Differential Neutrophil Count: Geometric Means and 95% CI by timepoint and challenge (baseline, 26h LPS Lobe, 26h Saline Lobe) and treatment group | | HR [1], SAC [1] | | |
| 2.11 | Evaluable | PD_F3 | BAL Differential Neutrophil Count: Participant Profiles of Baseline (2h) to 26h by Challenge and Treatment Group | Use participant attributes map so each subject has specific marker, line colour, pattern to track participant between plots. | HR [1], SAC [1] | | |
| Pharmac | odynamic: Fi | gures | | | |
|---|---|---|---|---|---|
| No. | Populati<br>on | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.12 | Evaluable | PD_F4 | <b>BAL Differential Neutrophil Count</b> : Point Estimates and 95% Credible Intervals | Page to include 3 column panels. 1st: (Back-transformed) treatment group predictions, 2nd: Treatment group differences, 3rd: Percentage reduction ('745 c.f. Pbo). | HR [1], SAC [1] |
| 2.13 | Evaluable | PD_F5 | BAL Differential Neutrophil Count: Posterior Distribution Density Plots from the Analysis | 3 pages in total. Page 1: posteriors for separate treatment groups. Page 2: posterior for absolute difference (GSK2798745 c.f. placebo) Page 3: posterior for percentage reduction (GSK2798745 c.f. placebo) | HR [1], SAC [1] |
| Explorato | ory BAL Biom | narkers | | | |
| 2.14 | Evaluable | PD_F1 | <b>Exploratory BAL Biomarkers (excluding WBCs):</b> Geometric Means and 95% CI of by timepoint and challenge (baseline, 26 h LPS Lobe, 26 h Saline Lobe) and treatment group | One page per biomarker. | SAC [1] |
| 2.15 | Evaluable | PD_F3 | Exploratory BAL Biomarkers (excluding WBCs): Participant Profiles of Baseline (2h) to 26h by Challenge and Treatment Group | One page per biomarker. Use participant attributes map so each subject has specific marker, line colour, pattern to track participant between plots. | SAC [1] |
| 2.16 | Evaluable | PD_F4 | Exploratory BAL Biomarkers (excluding WBCs): Point Estimates and 95% Credible Intervals from the Analyses | One page per biomarker. Page to include 3 column panels. 1st: (Back-transformed) treatment group predictions, 2nd: Treatment group differences, 3rd: Percentage reduction ('745 c.f. Pbo). | SAC [1] |

| Pharmac | Pharmacodynamic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Populati<br>on | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.17 | Evaluable | PD_F5 | Exploratory BAL Biomarkers (excluding WBC): Posterior Distribution Density Plots from the Analyses | 3 pages per analyte. Page 1: posteriors for separate treatment groups. Page 2: posterior for absolute difference (GSK2798745 c.f. placebo) Page 3: posterior for percentage reduction (GSK2798745 c.f. placebo). Treatment comparison for percentage change should be expressed as an increase/reduction depending on desired treatment direction for the specific analyte e.g. % reduction/increase 745 c.f. placebo. | SAC [1] |
| 2.18. | Evaluable | PD_F1 | BAL White Blood Cell Types (Totals and Differentials, except Neutrophils): Geometric Means and 95% CI by timepoint and challenge (baseline, 26 h LPS Lobe, 26 h Saline Lobe) and treatment group | One page per biomarker. | SAC [1] |
| 2.19. | Evaluable | PD_F3 | BAL White Blood Cell Types (Totals and Differentials, except Neutrophils): Participant Profiles of Baseline (2h) to 26h by Challenge and Treatment Group | One page per biomarker. Use participant attributes map so each subject has specific marker, line colour, pattern to track participant between plots. | SAC [1] |
| 2.20. | Evaluable | PD_F4 | BAL White Blood Cell Types (Totals and Differentials, except Neutrophils): Point Estimates and 95% Credible Intervals from the Analyses | One page per biomarker. Page to include 3 column panels. 1st: (Back-transformed) treatment group predictions, 2nd: Treatment group differences, 3rd: Percentage reduction ('745 c.f. Pbo). | SAC [1] |

| Pharmac | odynamic: Fi | gures | | | |
|---|---|---|---|---|---|
| No. | Populati<br>on | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.21 | Evaluable | PD_F5 | BAL White Blood Cell Types (Totals and Differentials, except Neutrophils): Posterior Distribution Density Plots from the Analyses | 3 pages per analyte. Page 1: posteriors for separate treatment groups. Page 2: posterior for absolute difference (GSK2798745 c.f. placebo) Page 3: posterior for percentage reduction (GSK2798745 c.f. placebo). Treatment comparison for percentage change should be expressed as an increase/reduction depending on desired treatment direction for the specific analyte e.g. % reduction/increase 745 c.f. placebo. | SAC [1] |
| BAL Pha | rmacodynam | ic/Biomarker adju | sted for Dilution Factor | | |
| 2.22 | Evaluable | PD_F1 | All BAL Biomarkers adjusted for Dilution Factor: Geometric Means and 95% CI by timepoint and challenge (baseline, 26 h LPS Lobe, 26 h Saline Lobe) and treatment group | Conditional Output. Urea-corrected. One page per biomarker. | SAC [1] |
| 2.23 | Evaluable | PD_F3 | All BAL Biomarkers adjusted for Dilution Factor: Participant Profiles of Baseline (2h) to 26h by Challenge and Treatment Group | Conditional Output. Urea-corrected. One page per biomarker. Use participant attributes map so each subject has specific marker, line colour, pattern to track participant between plots. | SAC [1] |

| Pharmaco | odynamic: Fi | gures | | | |
|---|---|---|---|---|---|
| No. | Populati<br>on | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.24 | Evaluable | PD_F4 | All BAL Biomarkers adjusted for Dilution Factor: Point Estimates and 95% Credible Intervals from the Analyses | Conditional Output. Urea-corrected. One page per biomarker. Page to include 3 column panels. 1st: (Back-transformed) treatment group predictions, 2nd: Treatment group differences, 3rd: Percentage reduction ('745 c.f. Pbo). | SAC [1] |
| 2.25 | Evaluable | PD_F5 | All BAL Biomarkers Corrected for Dilution Factor: Posterior Distribution Density Plots from the Analyses | Conditional Output. Urea-corrected. 3 pages per analyte. Page 1: posteriors for separate treatment groups. Page 2: posterior for absolute difference (GSK2798745 c.f. placebo) Page 3: posterior for percentage reduction (GSK2798745 c.f. placebo). Treatment comparison for percentage change should be expressed as an increase/reduction depending on desired treatment direction for the specific analyte e.g. % reduction/increase 745 c.f. placebo. | SAC [1] |
| Explorato | ry Blood Bio | markers | | | |
| 2.26 | Evaluable | PD_F1 | <b>Exploratory Blood Biomarkers:</b> Geometric Means and 95% CI by timepoint and treatment group | One page per biomarker. | SAC [1] |

| Pharmacodynamic: Figures | | | | | |
|---|---|---|---|---|---|
| No. | Populati<br>on | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.27 | Evaluable | PD_F7 | <b>Exploratory Blood Biomarkers:</b> Participant Time Profiles by Treatment Group | One page per biomarker. Use participant specific attributes map. Use discrete x-axis scale so timepoints 2h and 3h are distinguishable. For each biomarker decided on y-axis on case-by-case basis. | SAC [1] |
| 2.28 | Evaluable | PD_F6 | <b>Exploratory Blood Biomarkers:</b> Time Profiles of Adjusted Posterior Medians and 95% Credible Intervals. | 3 pages per biomarker. Page 1: Separate profiles for each treatment group. Page 2: Profile for absolute difference treatment comparison. Page 3: Treatment comparison as percentage change. | SAC [1] |
| 2.29 | Evaluable | PD_F5 | Exploratory Blood Biomarkers: Posterior Distribution Density Plots from the Analyses for each Timepoint | 6 pages per biomarker: First 4 pages: posterior for each treatment group on same page, 1 page per timepoint. Page 5: Analyte response absolute difference (GSK2798745 c.f. placebo) for all timepoints. Page 6: Analyte response percentage reduction (GSK2798745 c.f. placebo) for all timepoints. | SAC [1] |

# 12.11.7. Safety Tables

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events (AEs) | | | | |
| 3.1. | All Subjects | AE1 | Summary of All Adverse Events by System Organ Class and Preferred Term | ICH E3 | SAC [1] |
| 3.2. | All Subjects | AE1 | Summary All Drug-Related Adverse Events by System Organ Class and Preferred Term/by Overall Frequency | ICH E3 | SAC [1] |
| Serious | and Other Sig | nificant Adverse I | Events | | |
| 3.3. | All Subjects | AE16 | Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Participants and Occurrences) | FDAAA, EudraCT | SAC [1] |
| 3.4. | All Subjects | AE1 | Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study by System Organ Class and Preferred Term | IDSL | SAC [1] |
| Laborat | tory: Chemistry | 1 | | | |
| 3.5. | All Subjects | LB1 | Summary of Chemistry Changes from Baseline | ICH E3 | SAC [1] |
| Laborat | tory: Haematol | ogy | | | |
| 3.6. | All Subjects | LB1 | Summary of Haematology Changes from Baseline | ICH E3 | SAC [1] |
| Laborat | tory: Urinalysis | | | | |
| 3.7. | All Subjects | LB1 | Summary of Urine Concentration Changes from Baseline | ICH E3 | SAC [1] |
| 3.8. | All Subjects | UR3 | Summary of Urinalysis Dipstick Results | ICH E3 | SAC [1] |
| Laborat | tory: Hepatobili | iary (Liver) | | | |
| 3.9. | All<br>Subjects | LIVER1 | Summary of Liver Monitoring/Stopping Event Reporting | IDSL | SAC [1] |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| ECG | , | | | | |
| 3.10. | All<br>Subjects | EG1 | Summary of ECG Findings | IDSL | SAC [1] |
| 3.11. | All Subjects | EG2 | Summary of Change from Baseline in ECG Values by Visit | IDSL | SAC [1] |
| 3.12. | All Subjects | SAFE_T4 | Summary of Number of Participants with Maximum ECG Values Meeting or Exceeding Pre-Specified Ranges of Concern by Category, Treatment and Timepoint. | | SAC [1] |
| Vital Sig | gns | | | | |
| 3.13. | All Subjects | VS1 | Summary of Change from Baseline in Vital Signs | ICH E3 Include body temperature, heart rate, blood pressure. | SAC [1] |
| Columb | oia Suicide Sev | erity Rating Scale | (C-SSRS) | | |
| 3.14. | All Subjects | CSSRS1<br>(SAFE_T1) | Summary of C-SSRS Suicidal Ideation or Behaviour | Include Placebo column. | SAC [1] |
| Laborat | tory: Other | | | | |
| 3.15. | All Subjects | SAFE_T2 | Summary of Faecal Occult Blood Test (FOBT) Data | | SAC [1] |
| 3.16. | All Subjects | LB1 | Summary of Cardiac Troponin (cTn) Changes from Baseline | | SAC [1] |
| 3.17. | All Subjects | LB1 | Summary of Coagulation Profile Changes from Baseline | | SAC [1] |
| Spirom | etry | | | <u> </u> | |
| 3.18. | All Subjects | SAFE_T3 | Summary of Spirometry Data | | SAC [1] |

# 12.11.8. Pharmacokinetic Tables

| Pharma | Pharmacokinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Plasma | PK Concentra | tion | | | • |
| 4.1. | PK | PKCT1 / PK01 | Summary of GSK2798745 Plasma Pharmacokinetic Concentration-Time Data (ng/mL) | | SAC [1] |
| 4.2. | PK | PKCT1 / PK01 | Summary of Metabolite GSK3526876 Plasma Pharmacokinetic Concentration-Time Data (ng/mL) | Conditional output. | SAC [1] |
| BAL P | Concentration | n | | | • |
| 4.3. | PK | PKCT1 / PK01 | Summary of GSK2798745 BAL 2h and 26h Concentration Data (ng/mL) | Not urea-corrected. | SAC [1] |
| 4.4. | PK | PKCT1 / PK01 | Summary of GSK2798745 BAL 2h and 26h Concentration Corrected for Dilution Factor Data (ng/mL) | Conditional output. Urea-corrected. | SAC [1] |
| Plasma | PK Parameter | S | | | • |
| 4.5. | PK | PKPT1 / PK03 | Summary of Derived GSK2798745 Plasma Pharmacokinetic Parameters | | SAC [1] |
| 4.6. | PK | PKPT3 / PK05 | Summary of Log-Transformed Derived GSK2798745 Plasma Pharmacokinetic Parameters | | SAC [1] |
| 4.7. | PK | PKPT1 / PK03 | Summary of Derived Metabolite GSK3526876 Plasma Pharmacokinetic Parameters | Conditional output. | SAC [1] |
| 4.8. | PK | PKPT3 / PK05 | Summary of Log-Transformed Derived Metabolite GSK3526876 Plasma Pharmacokinetic Parameters | Conditional output. | SAC [1] |

# 12.11.9. Pharmacokinetic Figures

| Pharma | Pharmacokinetic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Plasma | PK Concentra | tions | | | |
| 4.1. | PK | PKCF1P /<br>PK16a | Individual GSK2798745 Plasma Concentration-Time Plot (Linear and Semi-Log) | | SAC [1] |
| 4.2. | PK | PKCF2 / PK17 | Mean GSK2798745 Plasma Concentration-Time Plot (Linear and Semi-Log) | | SAC [1] |
| 4.3. | PK | PKCF3 / PK18 | Median GSK2798745 Plasma Concentration-Time Plot (Linear and Semi-Log) | | SAC [1] |
| 4.4. | PK | PKCF1P /<br>PK16a | Individual Metabolite GSK3526876 Plasma Concentration-Time Plot (Linear and Semi-Log) | Conditional output. | SAC [1] |
| 4.5. | PK | PKCF2 / PK17 | Mean Metabolite GSK3526876 Plasma Concentration-Time Plot (Linear and Semi-Log) | Conditional output. | SAC [1] |
| 4.6. | PK | PKCF3 / PK18 | Median Metabolite GSK3526876 Plasma Concentration-Time Plot (Linear and Semi-Log) | Conditional output. | SAC [1] |
| BAL P | Concentration | าร | | | |
| 4.7. | PK | PK_F1 | Individual Participant and Median BAL GSK2798745<br>Concentration-Time Plot | Not urea-corrected BAL concentration. PK_F1 is a loose example. One active treatment group in this study. Use participant-specific attributes map. | SAC [1] |
| 4.8. | PK | PK_F1 | Individual Participant and Median BAL GSK2798745 Concentration-Time Plot (Concentration Adjusted for Dilution Factor) | Conditional output. Urea-corrected BAL concentration. PK_F1 is a loose example. One active treatment group in this study. Use participant-specific attributes map. | SAC [1] |

| Pharma | Pharmacokinetic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| BAL an | d Plasma PK C | oncentrations | | | |
| 4.9. | Evaluable | PKPD_F1 | Scatter Plots of Plasma PK Parameters (C <sub>MAX</sub> , AUC <sub>0-26</sub> , C <sub>26</sub> ) v BAL GSK2798745 Concentrations (C <sub>2</sub> , C <sub>26</sub> ). | Only participants on active treatment. Page 1: Plasma C <sub>MAX</sub> v BAL C <sub>2</sub> . Page 2: Plasma AUC <sub>0-26</sub> v BAL C <sub>26</sub> Page 3: Plasma C <sub>26</sub> v BAL C <sub>26</sub> | SAC [1] |
| 4.10. | Evaluable | PKPD_F1 | Scatter Plots of Plasma PK Parameters (C <sub>MAX</sub> , AUC <sub>0-26</sub> , C <sub>26</sub> ) v<br>BAL GSK2798745 Concentrations (C <sub>2</sub> , C <sub>26</sub> ). <b>BAL</b><br><b>Concentrations Adjusted for Dilution Factor.</b> | Only participants on active treatment. Page 1: Plasma C <sub>MAX</sub> v BAL C <sub>2</sub> . Page 2: Plasma AUC <sub>0-26</sub> v BAL C <sub>26</sub> Page 3: Plasma C <sub>26</sub> v BAL C <sub>26</sub> | SAC [1] |

# 12.11.10. Pharmacokinetic / Pharmacodynamic Figures

| Pharma | Pharmacokinetic / Pharmacodynamic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK / PD | | | | | |
| 7.1. | Evaluable | PKPD_F1 | Scatter Plots of Plasma PK Parameters (AUC <sub>0-26</sub> , C <sub>26</sub> , C <sub>max</sub> ) v 26h BAL Total Protein. | Page 1: Plasma AUC <sub>0-26</sub> v 26h BAL Total<br>Protein<br>Page 2: Plasma C <sub>26</sub> v 26h BAL Total<br>Protein<br>Page 3: Plasma C <sub>MAX</sub> v 26h BAL Total<br>Protein | SAC [1] |
| 7.2. | Evaluable | PKPD_F1 | Plots of BAL GSK2798745 Concentrations v 26h BAL Total Protein | Page 1: BAL C <sub>2</sub> v 26h BAL Total Protein<br>Page 2: BAL C <sub>26</sub> v 26h BAL Total Protein | SAC [1] |

# 12.11.11. ICH Listings

| ICH: Lis | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | • |
| 1. | Screened | ES7 | Listing of Reasons for Screen Failure | Journal Guidelines | SAC [1] |
| 2. | Enrolled | ES2 | Listing of Reasons for Study Withdrawal | ICH E3 | SAC [1] |
| 3. | All Subjects | SD2 | Listing of Reasons for Study Treatment Discontinuation | ICH E3 | SAC [1] |
| 4. | All Subjects | BL1 | Listing of Participants for Whom the Treatment Blind was Broken | ICH E3 | SAC [1] |
| 5. | All Subjects | TA1 / CP_RD1x | Listing of Planned and Actual Treatments | IDSL | SAC [1] |
| Protoco | ol Deviations | | | | • |
| 6. | All Subjects | DV2 | Listing of Important Protocol Deviations | ICH E3 | SAC [1] |
| 7. | All Subjects | IE3 | Listing of Participants with Inclusion/Exclusion Criteria Deviations | ICH E3 | SAC [1] |
| Popula | tions Analysed | | | | • |
| 8. | All Subjects | SP3 | Listing of Participants Excluded from Any Population | ICH E3 | SAC [1] |
| Demog | raphic and Bas | eline Characterist | ics | | |
| 9. | Screened | DM2 | Listing of Demographic Characteristics | ICH E3 | SAC [1] |
| 10. | Screened | DM9 | Listing of Race | ICH E3 | SAC [1] |
| Prior a | Prior and Concomitant Medications | | | | |
| 11. | All Subjects | CP_CM3 | Listing of Concomitant Medications | IDSL | SAC [1] |

| ICH: Lis | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Exposu | re and Treatme | ent Compliance | | | |
| 12. | All Subjects | EX3 | Listing of Exposure Data | ICH E3 | SAC [1] |
| Advers | e Events | | | | |
| 13. | All Subjects | AE8CP | Listing of All Adverse Events | ICH E3 | SAC [1] |
| 14. | All Subjects | AE7 | Listing of Participant Numbers for Individual Adverse Events | ICH E3 | SAC [1] |
| 15. | All Subjects | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text | IDSL | SAC [1] |
| Serious | and Other Sig | nificant Adverse I | -<br>Events | | |
| 16. | All Subjects | AE8CPa | Listing of Fatal Serious Adverse Events | ICH E3 | SAC [1] |
| 17. | All Subjects | AE8CPa | Listing of Non-Fatal Serious Adverse Events | ICH E3 | SAC [1] |
| 18. | All Subjects | AE14 | Listing of Reasons for Considering as a Serious Adverse Event | ICH E3 | SAC [1] |
| 19. | All Subjects | AECP8 | Listing of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment | ICH E3 | SAC [1] |
| 20. | All Subjects | AECP8 | Listing of Other Significant Adverse Events | ICH E3 | SAC [1] |
| Hepato | biliary (Liver) | | | | |
| 21. | All Subjects | MH2 | Listing of Medical Conditions for Participants with Liver Stopping Events | IDSL | SAC [1] |
| 22. | All Subjects | SU2 | Listing of Substance Use for Participants with Liver Stopping Events | IDSL | SAC [1] |
| All Lab | oratory | | | | |
| 23. | All Subjects | LB5 | Listing of All Laboratory Data for Participants with Any Value of Potential Clinical Importance | ICH E3 | SAC [1] |
| 24. | All Subjects | LB5 | Listing of Laboratory Values of Potential Clinical Importance | | SAC [1] |

| ICH: Lis | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 25. | All Subjects | LB14 | Listing of Laboratory Data with Character Results | ICH E3 | SAC [1] |
| 26. | All Subjects | UR2A | Listing of Urinalysis Data for Participants with Any Value of Potential Clinical Importance | ICH E3 | SAC [1] |
| ECG | | | | | |
| 27. | All Subjects | EG3 | Listing of All ECG Values for Participants with Any Value of Potential Clinical Importance | IDSL | SAC [1] |
| 28. | All Subjects | EG3 | Listing of ECG Values of Potential Clinical Importance | IDSL | SAC [1] |
| 29. | All Subjects | EG5 | Listing of All ECG Findings for Participants with an Abnormal ECG Finding | IDSL | SAC [1] |
| 30. | All Subjects | EG5 | Listing of Abnormal ECG Findings | IDSL | SAC [1] |
| Vital Si | gns | | | • | |
| 31. | All Subjects | VS4 | Listing of All Vital Signs Data for Participants with Any Value of Potential Clinical Importance | IDSL | SAC [1] |
| 32. | All Subjects | VS4 | Listing of Vital Signs of Potential Clinical Importance | IDSL | SAC [1] |

# 12.11.12. Non-ICH Listings

| Non-IC | H: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Pharma | acodynamic | | | | |
| 33. | Evaluable | PD_L2 | Listing of BAL Total Protein Data | | IA1 [1], IA2 [1],<br>HR [1], SAC [1] |
| 34. | Evaluable | PD_L2 | Listing of BAL Total Protein Data Corrected for Dilution Factor. | Conditional Output. Urea-corrected. | SAC [1] |
| 35. | Evaluable | PD_L2 | Listing of BAL Neutrophil Data (Total and Percentage) | Percentage in brackets – change template accordingly. | HR [1] |
| 36. | Evaluable | - | <b>26h BAL Total Protein</b> : Raw SAS Output from the Primary Analysis | | IA1 [1], IA2 [1],<br>HR [1], SAC [1] |
| 37. | Evaluable | - | Sensitivity Analysis: 26 h BAL Total Protein including 26h Saline Lobe BAL Total Protein as a Covariate: Raw SAS Output from the Analysis | | SAC [1] |
| 38. | Evaluable | - | Sensitivity Analysis 26 h BAL Total Protein Excluding Participants with High Saline Lobe BAL Total Protein Level: Raw SAS Output from the Analysis | | SAC [1] |
| 39. | Evaluable | - | Exploratory Analysis: 26 h BAL Total Protein and Total Neutrophil Count: Raw SAS Output from the Multivariate Analysis | Conditional Output. | SAC [1] |
| 40. | Evaluable | - | 26h BAL Total Neutrophil Count: Raw SAS Output from the Analysis | | SAC [1] |
| 41. | Evaluable | - | 26 h BAL Differential Neutrophil Count: Raw SAS Output from the Analysis | | SAC [1] |
| 42. | Evaluable | - | Exploratory BAL Biomarkers (excluding WBC): Raw SAS Output from the Analyses | | SAC [1] |

| Non-IC | H: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 43. | Evaluable | - | <b>BAL White Blood Cell Types (Totals and Differentials):</b> Raw SAS Output from the Analyses | | |
| 44. | Evaluable | - | All Exploratory BAL Biomarkers Corrected for Dilution Factor: Raw SAS Output from the Analysis | Conditional Output. Urea-corrected. | SAC [1] |
| 45. | Evaluable | - | Exploratory Blood Biomarkers: Raw SAS Output from the Analysis | | SAC [1] |
| Safety | | | | | |
| 46. | All Subjects | SAFE_L1 | Listing of Spirometry Data of Potential Clinical Importance | | SAC [1] |
| 47. | All Subjects | CSSRS4<br>(SAFE_L2) | Listing of C-SSRS Suicidal Ideation or Behaviour Data | | SAC [1] |
| 48. | All Subjects | CSSRS5<br>(SAFE_L3) | Listing of C-SSRS Suicidal Behaviour Details | Production dependent on events occurring. | SAC [1] |
| 49. | All Subjects | SAFE_L4 | Listing of Abnormal Faecal Occult Blood Test (FOBT) Data | | SAC [1] |
| Interim | Analysis Spec | ific | | | |
| 50. | Evaluable | PD_L1 | Interim Analysis: Raw SAS output from predicting the probability of achieving end of study success | | IA1 [1], IA2 [1],<br>HR [1], SAC [1] |
| Pharma | acokinetic | | | | |
| 51. | PK | PKCL1P / PK07 | Listing of GSK2798745 Plasma Pharmacokinetic Concentration-<br>Time Data | | SAC [1] |
| 52. | PK | PKPL1P / PK13 | Listing of Derived GSK2798745 Primary and Secondary Pharmacokinetic Parameters | | SAC [1] |
| 53. | PK | PKCL1P / PK07 | Listing of Metabolite GSK3526876 Plasma Pharmacokinetic Concentration-Time Data | | SAC [1] |

| Non-ICI | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 54. | PK | PKPL1P / PK13 | Listing of Derived Metabolite GSK3526876 Primary and Secondary Pharmacokinetic Parameters | | SAC [1] |
| 55. | PK | PKCL1P / PK07 | Listing of GSK2798745 BAL Pharmacokinetic Concentration-<br>Time Data | Not urea-corrected. | SAC [1] |
| 56. | PK | PKCL1P / PK07 | Listing of GSK2798745 BAL Pharmacokinetic Concentration-<br>Time Data <b>Adjusted for Dilution Factor</b> | Conditional output. Urea-corrected. | SAC [1] |

12.12. Appendix 12: Example Mock Shells for Data Displays

Example: PD\_T1 Page 1 of n

Protocol: 207464
Population: Evaluable

Table 2.1
Summary of BAL Total Protein by Timepoint (Baseline (2 h) and 26 h), Lung Lobe (LPS and Saline Challenge) and Treatment Group

| Parameter | Treatment | Timepoint/Chall | N | n | Arithmetic<br>Mean | Arithmetic<br>95% CI of<br>Mean | Arithmetic<br>SD | Median | Min | Max |
|---|---|---|---|---|---|---|---|---|---|---|
| BAL Total<br>Protein<br>(ug/mL) | Placebo | Baseline (2 h) | 30 | 30 | 92.07 | (76.647,<br>107.49) | 41.30 | 84.07 | 33.15 | 190.94 |
| | | LPS (26 h) | 30 | 30 | 290.39 | (214.00,<br>366.79) | 204.59 | 245.46 | 69.50 | 1113.5 |
| | | Saline (26 h) | 30 | 30 | 115.20 | (105.48,<br>124.92) | 26.02 | 111.34 | 65.68 | 167.58 |
| | GSK2798745 | Baseline (2 h) | 30 | 30 | 91.04 | (81.026,<br>101.06) | 26.83 | 90.58 | 46.29 | 145.77 |
| | | LPS (26 h) | 30 | 30 | 150.50 | (123.49,<br>177.51) | 72.33 | 145.34 | 71.69 | 370.73 |
| | | Saline (26 h) | 30 | 30 | 100.09 | (85.923,<br>114.26) | 37.94 | 90.11 | 45.34 | 194.93 |

Example: PD \_T1 Page 1 of n

Protocol: 207464
Population: Evaluable

Table 2.1 (continued)
Summary of BAL Total Protein by Timepoint (Baseline and 26 h), Lung Lobe (LPS and Saline Challenge) and Treatment Group

| Parameter | Treatment | Timepoint/Chall | N | n | Geometric<br>Mean | 95% CI of<br>Geometric<br>Mean | SD Logs |
|---|---|---|---|---|---|---|---|
| BAL Total<br>Protein<br>(ug/mL) | Placebo | Baseline | 30 | 30 | 93.81 | (58.657,<br>160.33) | 0.29 |
| | | LPS (26 h) | 30 | 30 | 248.80 | (95.136,<br>458.63) | 0.48 |
| | | Saline (26 h) | 30 | 30 | 95.15 | (44.451,<br>182.50) | 0.44 |
| | GSK2798745 | Baseline | 30 | 30 | 86.07 | (52.140,<br>129.92) | 0.30 |
| | | LPS (26 h) | 30 | 30 | 200.01 | (85.715,<br>402.44) | 0.51 |
| | | Saline (26 h) | 30 | 30 | 99.37 | (60.871,<br>142.52) | 0.30 |

Example: PD\_T2
Protocol: 207464

Page x of x

Population: Evaluable Data as of xx-xxx-xxxx

Table 2.3 (cont.)

| Endpoint/Analyte | Treatment | Item | n | Median | SD | 95% CrI |
|---|---|---|---|---|---|---|
| Total Protein | Placebo | Raw Baseline | Х | xxxxx | XXXX | (xxxx, xxxx) |
| | GSK2798745 | Raw Baseline | Х | xxxxx | xxxx | (xxxx, xxxx) |
| | N/a | Baseline Value used in Statistical Modelling | | xxxxxx | | |

Example: PD\_T2 (continued)

Protocol: 207464

Page x of x

Population: Evaluable Data as of xx-xxx-xxxx

Table 2.3 (cont.)

| Response/Analyte | Treatment | n | Median | SD | 95% CrI | 75% CrI | MCSE/SD |
|---|---|---|---|---|---|---|---|
| 26 h Total Protein | Placebo | Х | xxxxx | XXXXX | (xxxxx, xxxxx) | (xxxxx, xxxxx) | xxxxx |
| | GSK2798745 | Х | XXXXX | XXXXX | (xxxxx, xxxxx) | (xxxxx, xxxxx) | XXXXX |

Example: PD\_T2 (continued)

Protocol: 207464

Page x of x

Population: Evaluable Data as of xx-xxx-xxxx

Table 2.3 (cont.)

| Endpoint/Analyte | Comparison | Median | SD | 95% CrI | 75% CrI | MCSE/SD |
|---|---|---|---|---|---|---|
| 26 h Total Protein | Absolute Difference (Active - Placebo) | XXXXX | xxxxx | (xxxxx, xxxxx) | (xxxxx, xxxx) | xxxx |
| | Percentage Reduction (Active cf. Placebo) | xxxxx | xxxxx | (xxxxx, xxxxx) | (xxxxx, xxxx) | xxxx |

Example: PD\_T2 (continued)

Protocol: 207464

Page x of x

Population: Evaluable Data as of xx-xxx-xxxx

Table 2.3 (cont.)

| Response | Comparison | Posterior Probability Statement | Value |
|---|---|---|---|
| 26 h Total Protein | Median Percentage Change (Active cf. Placebo) | At least a 75% mean reduction (Active c.f. Placebo) | 0.002 |
| | | At least a 50% mean reduction (Active c.f. Placebo) | 0.221 |
| | | At least a 25% mean reduction (Active c.f. Placebo) | 0.522 |
| | | At least a 10% mean reduction (Active c.f. Placebo) | 0.721 |
| | | Any mean reduction (Active c.f. Placebo) | 0.952 |
| | | Any mean increase (Active c.f. Placebo) | 0.048 |
| | | At least a 10% mean increase (Active c.f. Placebo) | 0.030 |
| | | At least a 25% mean increase (Active c.f. Placebo) | 0.018 |
| | | At least a 50% mean increase (Active c.f. Placebo) | 0.002 |
| | | At least a 75% mean increase (Active c.f. Placebo) | 0.000 |

Example: PD\_F1
Protocol: 207464
Population: Evaluable


Figure 2.10
Boxplots of Total Protein by Timepoint/Challenge and Treatment Group




Protocol: 207464
Population: Evaluable

Figure 2.73
Scatter Plot of 26 Total Protein v 26h Total Neutrophil in the LPS Challenged Lobe

#### 207464 Planning: Scatter plot of 26h Total Protein v 26h Total Neutrophil in the LPS Challenged Lobe



Note: correlation is rho value taken from unstructured variance-covariance matrix in multivariate analysis


Protocol: 207464 Population: Evaluable

Figure 2.12
Participant Profiles of Baseline (2h), LPS lobe (26h) and Saline Lobe (26h) BAL Total Protein by Treatment Group



Example: PD \_F4 Protocol: 207464 Population: Evaluable Page 1 of n

Table 2.13
Total Protein Point Estimates and 95% Highest Posterior Density Intervals from the Primary Analysis



Example: PD\_F5
Protocol: 207464
Population: Evaluable


Figure 2.14
Total Protein Posterior Density Plots from the Primary Analysis




Figure 2.83
Time Profiles of Adjusted Posterior Medians and 95% Credible Intervals for Blood Total Protein




207464

Example: PD \_F6 (continued)

Figure 2.83 (continued)




Figure 2.82
Participant Time Profiles of \*\*BLOOD BIOMARKER\*\* by Treatment Group



Example: PD\_L1 Page 1 of n

Protocol: 207464
Population: Evaluable

Listing 39
Raw SAS Output from Predicting the Probability of Achieving End of Study Success

| Success | Frequency<br>(Number of<br>Complete Studies) | Interim<br>Posterior<br>Predictive<br>Probability |
|---|---|---|
| Yes | 7602 | 0.76 |
| No | 2398 | 0.24 |

Note: End of Study Success Definition: Posterior Probability (% reduction Active compared to Placebo) ≥ 0.95

EXAMPLE CSSRS1 (SAFE T1) Protocol: GSK123456

 Population: All Subjects

Table X Summary of Participants with C-SSRS Suicidal Ideation or Behaviour during Treatment

| | | atment A<br>N=78) | | |
|---|---|---|---|---|
| Number of participants with at least one on-treatment C-SSRS assessment | 77 | | 78 | |
| Suicidal Ideation or Behaviour (1-10) Any event | 28 | (36%) | 34 | (44%) |
| Suicidal Ideation (1-5) Any suicidal ideation 1 - Passive: Wish to be dead 2 - Active: Non-specific (no method, intent, 3 - Active: Method, but no intent or plan 4 - Active: Method and intent, but no plan 5 - Active: Method, intent, and plan | 9<br>plan) 6<br>6<br>6 | (8%)<br>(8%) | 11<br>8<br>8<br>8 | (14%)<br>(10%)<br>(10%)<br>(10%) |
| Suicidal Behaviour (6-10) Any suicidal behaviour 6 - Preparatory acts or behaviour 7 - Aborted attempt 8 - Interrupted attempt 9 - Non-fatal actual suicide attempt 10 - Completed suicide | 9<br>6<br>6<br>6 | (36%)<br>(12%)<br>(8%)<br>(8%)<br>(8%)<br>(8%) | 11<br>8<br>8<br>8 | (14%)<br>(10%)<br>(10%) |
| Self-Injurious Behaviour, no suicidal attempt | 6 | (8%) | 8 | (10%) |

Note: Percentages are based on the number of participants with at least one on-treatment C-SSRS assessment. For behaviour, the numbers of participants (n) are those with the specified behaviour at least once during treatment. For ideation, n refers to the number whose maximum ideation at any on-treatment assessment is the specified ideation. Participants may have more than one type of suicidal ideation or behavior. USER ID: directory/ program.sas DDMMMYYYY HH:MM


# CONFIDENTIAL

Example: SAFE\_T2
Protocol: 207464

Population: All Subjects

Table 3.15 Summary of Faecal Occult Blood Test (FOBT) Data

| Parameter | Treatment | Timepoint/Chall | N | n | Number of<br>Positive<br>Results |
|---|---|---|---|---|---|
| Haemoglobin<br>(ng/ml) | Placebo | Screening | 30 | 30 | 0 |
| | | Follow-up | 30 | 30 | 1 |
| | GSK2798745 | Screening | 30 | 30 | 0 |
| | | Follow-up | 30 | 30 | 3 |


# CONFIDENTIAL

Example: SAFE\_T3
Protocol: 207464

Population: All Subjects

Table 3.17 Summary of Spirometry Data

| Treatment | Visit | Planned<br>Relative<br>Timepoi<br>nt | N | n | PFT<br>(Units) | Mean | 95% CI | Mean<br>%<br>Pred<br>FEV1<br>(L) | 95% CI | Mean<br>FEV1/<br>FVC<br>Ratio | 95% CI | # Participant s with % Pred FEV1 < 80% | # Participant s with % FEV1/FVC Ratio < 70% |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Placebo | Screening | Screenin<br>g | 30 | 29 | FEV1 (L) | 3.552 | 3.213, 3.901 | 82.44 | 76.72, 88.90 | | | 2 | |
| | | | 30 | 29 | FVC (L) | | | | | 5.505 | 5.212, 5.987 | | 3 |
| | Day -1 | Day -1 | | | FEV1 (L) | | | | | | | | |
| | | _ | | | FVC (L) | | | | | | | | |
| | Day 1 | Pre-dose | | | FEV1 (L) | | | | | | | | |
| | | | | | FVC (L) | | | | | | | | |
| | Day 1 | 6 h | | | FEV1 (L) | | | | | | | | |
| | | | | | FVC (L) | | | | | | | | |
| | Day 2 | 25.5 h | | | FEV1 (L) | | | | | | | | |
| | | | | | FVC (L) | | | | | | | | |
| | Day 2 | 30 h | | | FEV1 (L) | | | | | | | | |
| | | | | | FVC (L) | | | | | | | | |
| | Day 8 | Day 8 | | | FEV1 (L) | | | | | | | | |
| | | | | | FVC (L) | | | | | | | | |

Example: SAFE\_T4

Protocol: IPC103711


Population: All Subjects

Table 12.6

Summary of Number of Participants with Maximum ECG Values meeting or exceeding Pre-specified Ranges of concern by Category, Treatment and Timepoint

Timepoint = Screening Visit

| | Placebo<br>(N=12) | 066 25mcg QD (N=13) | 066 87.5mcg QD (N=12) |
|---|---|---|---|
| QTCB | | | |
| n | 12 | 13 | 12 |
| >450 to <480 | 1 (8%) | 4 (31%) | 6 (50%) |
| >=480 to <500 | 0 | 0 | 0 |
| >=500 | 0 | 0 | 0 |
| QTCF | | | |
| n | 12 | 13 | 12 |
| >450 to <480 | 0 | 0 | 0 |
| >=480 to <500 | 1 (8%) | 0 | 0 |
| >=500 | 0 | 0 | 0 |

Page 17 of 19

#### CONFIDENTIAL

EXAMPLE SAFE\_L1
Protocol: IPC103711

Protocol: IPC103/11
Population: All Subjects

Listing 17
Listing of Spirometry Data

| | | | | | 1 | | | | | 0 | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Subi | . Treatment | Visit | Planned<br>Relative<br>Time | Date/<br>Time | | | | | Normal | % Predicted Normal FEV1 [1] | FVC |
| PPC | 066<br>87.5mcg QD | | SCREENING | 10MAR2008/<br>10:55 | FEV1(L) | 5.07 | 5.01 | 5.1 5.1 | 5.041 | 101.172 | |
| | J - | | | | FVC(L) | 6.4 | 6.39 | 6.48 6.48 | | | 0.79 |
| | | DAY 1 | PRE-DOSE | PPD /<br>8:24 | FEV1(L) | | | 5.38 | | | |
| | | DAY 7 | PRE-DOSE | PPD / 7:58 | FEV1(L) | 5 | | 5 | | | |
| | | | POST-BRONCH | | FEV1(L) | 5.06 | | 5.06 | | | |
| | | DAY 8 | POST-BRONCH | PPD<br>14:22 | FEV1(L) | 5.29 | | 5.29 | | | |
| | 066<br>87.5mcg QD | | SCREENING | 01APR2008/<br>10:41 | FEV1(L) | 4.18 | 4.22 | 4.37 4.37 | 4.496 | 97.202 | |
| | _ | | | | FVC(L) | 5.76 | 5.8 | 5.99 5.99 | | | 0.73 |
| | | DAY 1 | | <b>PPD</b> 7:57 | FEV1(L) | 4.43 | | 4.43 | | | |
| | | DAY 7 | PRE-DOSE | PPD<br>8:04 | FEV1(L) | 4.38 | | 4.38 | | | |
| | | | POST-BRONCH | | FEV1(L) | 4.2 | | 4.2 | | | |
| | | DAY 8 | POST-BRONCH | | FEV1(L) | 4.31 | | 4.31 | | | |

[1] Values have been recalculated from raw data PPD

EXAMPLE CSSRS4 (SAFE L2)

2019N394925\_00 207464

Protocol: GSK123456 

Population: All Subjects

#### 

Treatment: Treatment A

| | | | | l Ideati | ion (1-5 | ) | S | Suicidal | Behaviou | ır (6-10) | | Non- |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Visit/ | (1) | (2)<br>Non- | (3) | | (5) | | (7) | (8) | (9)<br>Non- | | Suic. |
| Centre | Evaluation/ | Wish | spec. | With- | (4) | With | (6) | Abor- | Inter- | fatal | (10) | Self- |
| ID/ | Assessment | to | Sui- | out | With- | Plan | Prep. | ted | rupted | Actual | Comp. | Injur- |
| Sub- | Date/ | be | cidal | In- | out | and | Acts/ | At- | At- | At- | sui- | ious |
| ject | Study Day | Dead | Thoughts | tent | Plan | Intent | Beh. | tempt | tempt | tempt | cide | Beh. |
| PPD | Visit 2<br>(Baseline)/<br>Lifetime/<br>PPD<br>-14 | Yes | Yes | Yes | No | No | No | No | No | No | No | No |
| | Visit 2<br>(Baseline)/<br>Current<br>History/<br>PPD<br>-14 | Yes | Yes | No | No | No | | | | | | |
| | VISIT 7 (Week 20)/ Since last visit/ PPD 140 | Yes | Yes | No | Yes | No | No | No | Yes | No | No | No |
| | Visit 2<br>(Baseline)/<br>Lifetime /<br>PPD<br>-15 | No | Yes | Yes | No | No | No | No | No | No | No | No |

Note: The current history period is within the past XX months. If a participant has a lifetime evaluation shown, but not a current history evaluation, this indicates that the participant's most severe suicidal ideation occurred during the current history period. If the participant had an actual suicide attempt which was not a completed suicide, it is considered as (9) Non-fatal actual attempt.

USER ID: directory/program.sas DDMMMYYYY HH:MM

EXAMPLE CSSRS5 (SAFE L3)

# 2019N394925\_00 207464

Protocol: GSK123456 Page 1 of n

Population: e.g., All Subjects, Safety

Listing X

Listing of C-SSRS Suicidal Behaviour Details

Treatment: Treatment A

| Centre<br>ID/<br>Subject | Visit/<br>Evaluation/<br>Assessment<br>Date/<br>Study Day | Suicidal<br>Behaviour/<br>Number of<br>Events | Description | Actual<br>Attempt<br>Type | If Actual Attempt: Date/ Actual Lethality/ Potential Lethality | Com- pleted Sui- cide? | Date of Most<br>Recent<br>Behavior [1] |
|---|---|---|---|---|---|---|---|
| PPD | Visit 2<br>(Baseline)/<br>Lifetime/<br>PPD<br>-14 | Actual<br>Attempt/<br>3 | Subject PPD<br>PPD | Most<br>recent | 10FEB2005/ No or very minor physical damage/ Behaviour not likely to result in injury | | |
| | | | | Most<br>lethal | 10FEB2002/<br>Minor physical<br>damage/ | | |
| | | | | Initial/<br>First | 10JAN2002/<br>No or very minor<br>physical damage/<br>Behaviour not likely<br>to result in injury | | |
| | | Inter-<br>rupted<br>Attempt/<br>1 | Subject was prevented from PPD | | | | FEB2002 |

[1] This column relates to suicidal behaviour other than actual attempts, for screening/baseline only.

USER ID: directory/program.sas DDMMMYYYY HH:MM

2019N394925\_00 207464

Example: SAFE\_L4 Page 1 of n

Listing 41
Listing of Abnormal Faecal Occult Blood Test (FOBT) Data

| Treatment | Pa | rticipant | Visit | Date | Time | Haemoglobin<br>Value (ng/ml) |
|---|---|---|---|---|---|---|
| Placebo | | PPD | Screening | 04APR2018 | 08:09 | |
| | | | Follow-up | 17APR2018 | 09:09 | |
| | | | Screening | 06APR2018 | 10:09 | |
| | | | Follow-up | 19APR2018 | 11:09 | |
| GSK2798745 | | | Screening | 03APR2018 | 12:09 | |
| | | | Follow-up | 18APR2018 | 13:09 | |
| | | | Screening | 05APR2018 | 14:09 | |
| | | | Follow-up | 120APR2018 | 15:09 | |

Example: PK\_F1 Page 1 of n

Protocol: 207464
Population: All Subjects

Figure 4.7 Individual Participant and Median BAL GSK2798745 Concentration-Time Plot



NOTE: For BAL Supernatant the median for the 26H timepoints are zero due to majority of the values being assigned as NQ.

Example: PKPD\_F1

Protocol: 207464 Population: Evaluable Page 1 of n



Example: PD\_L2
Protocol: 207464

Protocol: 20/464
Population: Evaluable

Page 1 of n Data as of XX-XXX-2018

Listing 1

Listing of BAL Total Protein Data

Treatment: Placebo

Analyte: Total Protein (pg/ml)

| | | | 2h Analyte | 2h | 26h Saline <u>Lobe</u> | 26h LPS Lobe | 26h |
|---|---|---|---|---|---|---|---|
| Subject | Baseline (2 <u>h)</u><br>date/time | 26h date/<br>time | Concn BAL<br>(pg/ml) | Concn<br>Vol (ml) | Analyte<br>(pg/ml) | BAL<br>(pg/ml) | WOL. (ml) |
| PPD | 01AUG2018/<br>09:45 | 02AUG2018/<br>09:50 | 168 | | 188 | 450 | |

PPD

Example AE2

Protocol: GSK123456 Page 1 of 12

Population: All Subjects

Table 6.2 Listing of Relationship between System Organ Class and Verbatim Text

| System Organ Class | Preferred Term | Verbatim Text |
|---|---|---|
| Blood and lymphatic system disorders | Lymphadenopathy | ENLARGED LYMPH NODE |
| Cardiac disorders | Palpitations<br>Tachycardia nos | HEART PALPITATION<br>TACHYCARDIA |
| Ear and labyrinth disorders | Cerumen impaction Ear pain Tinnitus | CLOGGED EARS WITH EAR WAX<br>EARACHES IN BOTH EARS<br>RIGHT EAR PAIN<br>RINGING IN RIGHT EAR |
| Eye disorders | Asthenopia Conjunctivitis Dry eye nos Eye redness Vision blurred | TIRED EYES BILATERAL ACUTE CONJUNCTIVITIS CONJUNCTIVITIS DRY EYES REDDENED EYES BLURRED VISION BLURRY VISION WORSENING OF BLURRED VISION |
| Gastrointestinal disorders | Abdominal pain nos<br>Abdominal pain upper | ABDOMEN PAIN MID-EPIGASTRIC AREA PAIN STOMACH ACHE STOMACH CRAMPS STOMACH PAIN |
| | Abdominal tenderness | LOCALIZED AREA OF TENDERNESS R<br>ABDOMEN<br>MILD TENDERNESS RIGHT LOWER<br>ABDOMINAL QUADRANT |
| | Constipation<br>Diarrhoea nos<br>Dry mouth<br>Dyspepsia | CONSTIPATION DIARRHEA DRY MOUTH DYSPEPSIA HEARTBURN |